## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for 200630: A randomised, double blind (sponsor unblinded), placebo controlled, single ascending dose study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a IV dose of GSK2831781 in healthy volunteers and patients with plaque psoriasis |
| <b>Compound Number</b> | : | GSK2831781 |
| <b>Effective Date</b> | : | 24-JAN-2018 |

# **Description:**

The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2014N192690\_11.

This RAP is intended to describe the safety, tolerability, pharmacodynamic and efficacy analyses required for the study.

This RAP will be provided to the study team members to convey the content of the reporting efforts, specifically Statistical Analysis Complete (SAC).

#### **RAP Authors:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Lead statistician (Immuno Inflammation, SPDS) | 23-JAN-18 | Email |
| (Lead author) Statistician (Immuno Inflammation, SPDS) | NA | NA |
| Director Clinical Pharmacology (Immuno Inflammation, CPMS) | 22-JAN-18 | Email |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Experimental Development Physician (Immuno Inflammation, Experimental Medicine Unit) | 23-JAN-18 | Email |
| Snr Experimental Medicine Scientist (Immuno Inflammation, Experimental Medicine Unit) | 23-JAN-18 | Email |
| Discovery Medicine Physician (Immuno Inflammation, Experimental Medicine Unit) | 23-JAN-18 | Email |
| Senior Scientific Investigator (Immuno Inflammation Experimental Medicine Unit) | 23-JAN-18 | Email |
| Translational Scientist (Immuno Inflammation, Experimental Medicine Unit) | 22-JAN-18 | Email |
| Director (GCSP) | 22-JAN-18 | Email |
| Data Quality Lead, CPSSO | 23-JAN-18 | Email |
| Clinical Development Manager (Dermatology and Immuno Inflammation, CPSSO) | 23-JAN-18 | Email |
| Associate Programmer (Immuno Inflammation, QSI) | 23-JAN-18 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|------------------------------------------------|-----------|-----------------|
| Statistics Director (II Clinical Statistics) | 23-JAN-18 | Email |
| Director Programming (II Clinical Programming) | 24-JAN-18 | Email |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | | | N | |
| | 1.1. | RAP AM | nendments | |
| 2. | SHMM | ARY OF | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | _ | s to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | bjectives and Endpoints | |
| | 2.3. | • | esign | |
| | 2.4. | | al Analyses | |
| | | | , | |
| 3. | PLAN | NED ANA | LYSES | 12 |
| | 3.1. | | Analyses | |
| | 3.2. | Final An | alyses | 13 |
| 4. | Λ N Ι Λ Ι \ | veie DOE | PULATIONS | 1.1 |
| 4. | 4 1 | | Deviations | |
| | 4.1. | FIOLOCOI | Deviations | 14 |
| 5. | CONS | IDERATION | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | | S | |
| | 5.1. | | reatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline | e Definitions | 15 |
| e | CTLIDY | | ATION ANALYSES | 17 |
| 6. | 5100 | Y POPUL | .ATION ANALYSES | 17 |
| 7. | SAFET | Y ANAL | YSES | 17 |
| | 7.1. | | Events Analyses | |
| | 7.2. | | Laboratory Analyses | |
| | 7.3. | | afety Analyses | |
| _ | | | | |
| 8. | | | ALYSES | |
| | 8.1. | | luration (only for HV) | |
| | | 8.1.1. | Endpoint / Variables | |
| | | 8.1.2. | Summary Measure | |
| | | 8.1.3.<br>8.1.4. | Population of Interest | |
| | | 0.1.4. | 8.1.4.1. Statistical Methodology Specification | |
| | 8.2. | Body Su | urface Area (only for PsO) | |
| | 0.2. | 8.2.1. | Endpoint / Variables | |
| | | 8.2.2. | Summary Measure | |
| | | 8.2.3. | Population of Interest | |
| | | 8.2.4. | Statistical Analyses / Methods | |
| | 8.3. | PASI-rel | lated endpoints (only for PsO) | |
| | | 8.3.1. | Endpoint / Variables | |
| | | 8.3.2. | Summary Measure | |
| | | 8.3.3. | Population of Interest | |
| | | 8.3.4. | Statistical Analyses / Methods | |
| | | | 8.3.4.1. Statistical Methodology Specification | |
| | 8.4. | | elated endpoints (only for PsO) | |
| | | 8.4.1. | Endpoint / Variables | |
| | | 8.4.2. | Summary Measure | 23 |


| 200630 |
|--------|

| | | 8.4.3. | Population of Interest | 23 |
|---|---|---|---|---|
| | | 8.4.4. | Statistical Analyses / Methods | 23 |
| | | | 8.4.4.1. Statistical Methodology Specification | |
| | 8.5. | PGA-rel | ated endpoints (only for PsO) | 23 |
| | | 8.5.1. | Endpoint / Variables | |
| | | 8.5.2. | Summary Measure | |
| | | 8.5.3. | Population of Interest | |
| | | 8.5.4. | Statistical Analyses / Methods | |
| 9. | PHAR | MACOKI | NETIC ANALYSES | 24 |
| | 9.1. | Drug Co | oncentration Measures | 24 |
| | 9.2. | | Pharmacokinetic Parameters | |
| | | 9.2.1. | Population of Interest | 25 |
| | | 9.2.2. | Statistical Methods | |
| 10. | PHAR | MACODY | YNAMIC AND BIOMARKER ANALYSES | 25 |
| | 10.1. | IHC para | ameters | 25 |
| | | 10.1.1. | Endpoint / Variables | 26 |
| | | 10.1.2. | Summary Measure | 27 |
| | | 10.1.3. | Population of Interest | 27 |
| | | 10.1.4. | Statistical Methods | |
| | | | 10.1.4.1. Statistical Methodology Specification | 28 |
| | 10.2. | Epiderm | nis thickness (only for PsO) | |
| | | 10.2.1. | Endpoint / Variables | |
| | | 10.2.2. | Summary Measure | |
| | | 10.2.3. | Population of Interest | |
| | | 10.2.4. | Statistical Methods | |
| | | | 10.2.4.1. Statistical Methodology Specification | 29 |
| | 10.3. | Other P | D parameters | |
| | | 10.3.1. | Endpoint / Variables | 29 |
| | | 10.3.2. | Summary Measure | 30 |
| | | 10.3.3. | Population of Interest | |
| | | 10.3.4. | Statistical Methods | 30 |
| | 10.4. | Transcri | ptomics (biopsy and blood) | 30 |
| | | 10.4.1. | Endpoint / Variables | 30 |
| | | 10.4.2. | Summary Measure | 31 |
| | | 10.4.3. | Population of Interest | 31 |
| | | 10.4.4. | Statistical Methods | 31 |
| 11. | PHAR | MACOKI | NETIC / PHARMACODYNAMIC ANALYSES | 32 |
| 4.0 | | | 0.17.7.4.1.1.1.7.0.7.0 | |
| 12. | IMMU | NOGENI | CITY ANALYSES | 32 |
| 40 | | OLA N.I. A N.I. | ALVOCO (DADT D) | 00 |
| 13. | BAYE | SIAN AN | ALYSES (PART B) | 33 |
| 4.4 | ٨٥٥٥ | NDICEC | | 25 |
| 14. | | | iv 1. Drotocal Defined Cabadula of Frants | |
| | 14.1. | | ix 1: Protocol Defined Schedule of Events | |
| | | 14.1.1. | , | |
| | | | Healthy volunteers (DTH subjects) | |
| | 440 | | Psoriasis patients | 39 |
| | 14.2. | | ix 2: Study Phases and Treatment Emergent Adverse | 4.4 |
| | | ⊏vents . | | 41 |


| | 14.2.1. | Study Phases for Concomitant Medication | 41 |
|--------|----------|----------------------------------------------------|----|
| | 14.2.2. | | |
| 14.3. | Appendix | x 3: A&R Data sets | |
| | 14.3.1. | Subject-Level Variables | |
| | | 14.3.1.1. ADA Status | 42 |
| | | 14.3.1.2. Treatment | 42 |
| 14.4. | Appendix | x 4: Data Display Standards & Handling Conventions | 43 |
| | 14.4.1. | Reporting Process | 43 |
| | 14.4.2. | Reporting Standards | 43 |
| | 14.4.3. | Reporting Standards for Pharmacokinetic | 44 |
| 14.5. | Appendix | x 5: Reporting Standards for Missing Data | 45 |
| | 14.5.1. | Handling of Missing Data | 45 |
| | | 14.5.1.1. Handling of Missing and Partial Dates | 45 |
| 14.6. | Appendix | x 6: Values of Potential Clinical Importance | |
| | 14.6.1. | Laboratory Values | |
| | 14.6.2. | ECG | |
| | 14.6.3. | Vital Signs | |
| 14.7. | | x 7: Pharmacokinetic/Pharmacodynamic Analyses | 48 |
| | 14.7.1. | Pharmacokinetic / Pharmacodynamic Dataset | |
| | | Specification | |
| | 14.7.2. | Pharmacokinetic / Pharmacodynamic Methodology | |
| 14.8. | | x 8: Abbreviations & Trade Marks | |
| | 14.8.1. | Abbreviations | |
| | 14.8.2. | Trademarks | |
| 14.9. | | x 9: List of Data Displays | |
| | 14.9.1. | Data Display Numbering | |
| | 14.9.2. | Mock Example Shell Referencing | |
| | 14.9.3. | Deliverables | |
| | 14.9.4. | Study Population Tables | |
| | 14.9.5. | Efficacy Tables | |
| | 14.9.6. | Efficacy Figures | |
| | 14.9.7. | Safety Tables | |
| | 14.9.8. | Safety Figures | |
| | 14.9.9. | Pharmacokinetic Tables | |
| | | Pharmacokinetic Figures | |
| | | Pharmacodynamic / Biomarker Tables | |
| | | Pharmacodynamic / Biomarker Figures | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 14.10. | Appendix | x 10: Example Mock Shells for Data Displays | 91 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol

# 1.1. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Plan_Study200630_Final_V1 [7-Nov-2017] | |
| Reporting and Analysis Pla | n_Study200630_Amendment_Final_V1 [23-Jan-2018] |
| Soluble LAG3 concentrations | Change from free and complex sLAG-3 to total sLAG-3 |
| Transcriptomics | Analyses included |
| PK / PD Dataset<br>Specification | Details removed as per current TMF guidelines, the specifications for these datasets will need to be in a separate document, which will reside in eTMF. |
| Minor updates | <ul> <li>Clarification of some outputs</li> <li>Added details for the Bayesian analyses</li> <li>Separate sections/outputs for IHC parameters and epidermis thickness</li> <li>Categories for ECG to match the protocol</li> </ul> |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| PK parameters to be derived include AUC(0-week4), Vss and MRT | <ul> <li>PK parameters AUC(0-<br/>week4), Vss and MRT will<br/>not be derived</li> </ul> | These parameters are not<br>relevant for the study/program<br>and/or a monoclonal antibody |
| Dose proportionality will be assessed using the power model | No statistical analysis (e.g. using a power model) will be performed | Interim analyses to support DEC meetings showed that the PK data is clearly non-linear (less than proportional increase in exposure with increasing dose), and hence a statistical analysis to test dose proportionality is redundant |
| Effect on free and GSK2831781<br>bound sLAG-3 concentrations | Total sLAG-3 concentrations will be used instead of free and complex sLAG-3 | The assays for free and complex sLAG-3 are not quantitative, and therefore a new assay to measure total sLAG-3 was developed. PK/PD modelling will be used to investigate the time course of |


| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan Rationale for Changes | |
| | | free and complex sLAG-3. |

# 2.2. Study Objectives and Endpoints

| Objectives | End | lpoints |
|---|---|---|
| Primary | Primary | |
| To assess the safety and tolerability of single IV doses of GSK2831781 in healthy | | Laboratory safety data (haematology, clinical chemistry, urinalysis) |
| volunteers and psoriasis patients. | • | Vital signs (blood pressure, heart rate, body temperature) |
| | • | 12-lead ECGs |
| | • | Adverse events |
| | • | Inflammatory cytokine levels |
| Secondary Objectives | | ondary Endpoints |
| To evaluate the pharmacology and clinical effect of a single IV dose of GSK2831781 in a DTH model in healthy volunteers. | • | Change from baseline (PPD 1st challenge) of induration diameter from re-challenge at 3 days post-dose Duration of induration in the re-challenge Change from baseline (PPD 1st challenge) of LAG-3+ cells in biopsies of re-challenged skin at 3 days post-dose, measured by IHC |
| To evaluate the pharmacology of a single IV dose of GSK2831781 in psoriasis patients. | | Change from baseline in LAG-3+ cells in lesional biopsies at Day 29 measured by IHC |
| To evaluate the pharmacokinetics of single IV doses of GSK2831781 in healthy volunteers and psoriasis patients. | | GSK2831781 PK parameters following single intravenous dose: AUC(0-∞), AUC(0-t), AUC(0-Week4), %AUCex, Cmax, tmax, tlast, CL, Vss, MRT, λz and t ½ when assessable |
| To evaluate the immunogenicity of GSK2831781 administered as a single IV dose in healthy volunteers and psoriasis patients. | • | Antibodies to GSK2831781 in serum |
| To evaluate the effect of a single IV dose of GSK2831781 on disease activity in psoriasis patients. | • | Change from baseline and actual PASI scores at Day 15, 29, 43, 85, 121 and follow-up |
| | • | Proportion of subjects who achieve ≥50% and ≥75% improvement from baseline in PASI score at Day 15, 29, 43, 85, 121 and follow-up (PASI 50 and PASI 75) |
| | | Change from baseline and actual PLSS scores at Day 15, 29, 43, 85, 121 and follow-up |
| | | Change from baseline and actual PGA scores at Day 15, 29, 43, 85 and 121 |
| | • | Proportion of subjects in each PGA score category at Day 15, 29, 43, 85 and 121 |
| | • | Proportion of subjects achieving PGA 0/1 and at least a 2-point improvement at Day 15, 29, 43, 85 and 121 |

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the effect of a single IV dose of GSK2831781 in psoriasis patients on biomarkers. | <ul> <li>Histopathological scoring of psoriatic lesional biopsies in<br/>subjects with psoriasis - Ki67, CD3 and epidermal thickness</li> </ul> |
| | <ul> <li>Transcriptomic analysis of psoriatic lesional biopsies in<br/>subjects with psoriasis</li> </ul> |
| To evaluate the effect of a single IV dose of GSK2831781 in healthy volunteers and psoriasis patients on pharmacodynamic biomarkers. | Proof of pharmacology biomarker endpoints may include, but not limited to, the following as data permit: • LAG-3 expression on different blood immune cell populations including T-cells • Transcriptomic profiling to assess mRNA levels in peripheral blood • Quantification of LAG-3 mRNA in whole blood • Inflammatory cytokine levels • sLAG-3 concentrations • NK cell CD16 receptor occupancy in whole blood • NK cell activation marker expression in whole blood |
| To explore the impact of pre-existing ADAs on the PK of GSK2831781 | <ul> <li>GSK2831781 PK parameters following single intravenous dose: AUC(0-∞), AUC(0-t), AUC(0-Week4), %AUCex, Cmax, tmax, tlast, CL, Vss, MRT, λz and t ½ when assessable</li> </ul> |

# 2.3. Study Design



#### **Overview of Study Design and Key Features**

#### Dosing

This is a dose escalation study, the planned dosing as per protocol is as below:

| Planned<br>Doses | Number of<br>subjects<br>randomised<br>(active:placebo) | Safety Follow-up<br>period to<br>progress to next<br>subjects/cohorts | PPD DTH<br>Challenge<br>if Healthy<br>volunteer/<br>Biopsy if<br>subject | Follow-up and end of exclusion of systemic immunosuppressives |
|---|---|---|---|---|
| Healthy Volui | nteers | | | |
| 0.0003mg/kg | 1:1 | 1:1 wait 28 days post-dose | No DTH | Day 29 ± 1 day<br>(28 days post-dosing) |
| 0.0015mg/kg | | | | Day 43 ± 1 day<br>(42 days post-dosing) |
| 0.0075mg/kg | 6:2 | 1:1 wait 48 hours post-dose | No DTH | Day 85 ± 2 days<br>(84 days post-dosing) |
| 0.04mg/kg | | 5:1 wait 28 days post-dose | | Day 147 ± 3 days<br>(146 days post-dosing) |
| 0.15mg/kg | 6:6 | 1:1 wait 48 hours<br>post-dose<br>5:5 wait 28 days<br>post-dose | DTH | Day 219 ± 7 days<br>(190 days post-dosing) |
| 0.15mg/kg* | 6:2 | 1:1 wait 48 hours<br>post-dose<br>5:1 wait 28 days<br>post-dose | No DTH | Day 189 ± 7 days<br>(190 days post-dosing) |

#### Notes:

- 1. Cohort with a DTH starts dosing on Day 29
- 2. DTH cohort at dose level 0.15mg/kg is in subjects with pre-existing ADA. All previous cohorts are in subjects without pre-existing ADA
- 3. Maximum dose for healthy volunteers may change based on emerging exposure

| Psoriasis pat | Psoriasis patients (Pre-existing ADA- and ADA +) | | | |
|---|---|---|---|---|
| 0.5mg/kg | 6:3 | 1:1 wait 48<br>hours post-dose<br>5:2 wait 28 days | Biopsy | 230 days post-dosing<br>± 7 days [no change<br>with amend #10] |
| 1.5mg/kg | | post-dose | | 183 days post-dosing<br>± 7† days (prior to<br>Amendment 10 was<br>270 days) |
| 5mg/kg | | | | 183 days post-dosing<br>± 7† days (prior to<br>Amendment 10 was<br>300 days) |

Note: All follow-up days may be increased or decreased during the study based on emerging data

† All subjects in Cohort 7 (0.5mg/kg) completed the day  $230 \pm 7$  follow up visit. Any subjects in Cohort 7 who have not had a 12-month surveillance visit when the amendment is approved should instead have a surveillance telephone call as soon as practically possible after the amendment is approved, rather than waiting to month 12 after dosing. Subjects in Cohort 8 (1.5mg/kg) who have already completed their follow up visit should also have a surveillance telephone call as soon as protocol amendment 10 is approved.

| Overview of Study Design and Key Features | |
|---|---|
| | Subjects in Cohort 8 (1.5mg/kg) and Cohort 9 (5mg/kg) who have not yet had a follow up visit when protocol amendment 10 is approved should have final assement, a combined follow up/surveillance visit at day 183 ± 7, or as soon as practically possible if they have already been monitored for longer than 183 ± 7 days after dosing. Subjects in Cohort 8 (1.5mg/kg) who have already completed their follow up visit should have their final assessment, a surveillance telephone call as soon as the protocol amendment is approved. |

# 2.4. Statistical Analyses

The primary objective is to determine the safety and tolerability of single IV doses of GSK2831781 in healthy volunteers and with mild to moderate psoriasis patients. There are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

| Interim<br>Analysis | Details (Protocol Defined) |
|---|---|
| Dose escalation | For Parts A and B of the study, review of safety, tolerability, available pharmacokinetic, DTH induration, available biomarker and PD for healthy volunteers or PASI and PLSS for psoriasis patients at the end of each cohort will be performed by DEC to aid decisions to proceed to higher dose strengths or to subjects with pre-existing ADA. This analysis can include review of individual subject data, summaries, graphical presentations and/or statistical analysis. |
| | Safety/tolerability data monitoring and the decision to proceed to the next dose level of GSK2831781 or to subjects with pre-existing ADA will be made by the DEC. |
| | The GSK Clinical Pharmacology Modeling and Simulation (CPMS) representative will extract PK data (including treatment information) from SMS2000 using unscrambled subject IDs. PK data will provide supporting evidence for each dose modification decision. Importantly, if the emerging PK data is significantly different from the predicted values, adjustment may have to be made to the planned doses. Dose modification decisions will take into account the emerging PK data, new PK prediction for the next dose and thus the expected safety cover for the next dose. |
| Interim 1 | <ul> <li>Formal unblinded interim analysis when the last subject in DTH cohort (cohort 5) has<br/>completed W4 visit. Data for healthy volunteers in cohorts 1-5 will be included.</li> </ul> |
| | The purpose of this interim analysis is to provide the project team and GSK stakeholders with key data to inform internal decision making, in order to plan future studies within the clinical development for the asset. |
| | There are no planned implications for the conduct of the study. |
| | Appropriate data summaries will be at the subject and treatment group level for key endpoints of interest and the circulation of results will be restricted to selected members of the project team and key GSK stakeholders. Results or discussions will |

| Interim<br>Analysis | Details (Protocol Defined) |
|---|---|
| | not be circulated to blinded staff involved in the conduct of the study at the sites. |
| Interim 2 | <ul> <li>Formal unblinded interim analysis will be conducted during part B. The PASI and<br/>PLSS will be evaluated when the last psoriasis patient in cohort 9 has completed D43<br/>visit, and the full interim 2 evaluation will be conducted after all patients have<br/>completed their day 85 visit. Data for healthy volunteers and psoriasis patients will be<br/>included.</li> </ul> |
| | <ul> <li>The purpose of this interim analysis is to provide the project team and GSK<br/>stakeholders with key data to inform internal decision making, in order to plan future<br/>studies within the clinical development for the asset.</li> </ul> |
| | There are no planned implications for the conduct of the study. |
| | <ul> <li>Appropriate data summaries will be at the subject and treatment group level for key endpoints of interest and the circulation of results will be restricted to selected members of the project team and key GSK stakeholders. Results or discussions will not be circulated to blinded staff involved in the conduct of the study at the sites.</li> </ul> |

# 3.2. Final Analyses

Final analyses will be reported when all subjects in all cohorts have completed their final scheduled visits (combined follow-up/surveillance visit or surveillance telephone call), and the following sequential steps have occurred:

- All subjects have completed the study as defined in the protocol.
- All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- All criteria for unblinding the randomisation codes have been met.
- Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Study Population |
| Safety | All randomized participants who received at least one dose of study treatment. | <ul><li>Study Population</li><li>Safety</li></ul> |
| | This population will be based on the treatment the subject actually received. | <ul><li>Efficacy</li><li>PD</li></ul> |
| | Note: Participants who were not randomized but received at least one dose of study treatment should be listed. | • lg |
| Pharmacokinetic (PK) | All participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values). | • PK |
| | This population will be based on the treatment the subject actually received. | |

Refer to Appendix 9 which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed, separately for healthy volunteers and psoriasis patients.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (30 September 2015 - version 2).

- Data will be reviewed and deviation will be finalised before freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A listing of all inclusion/exclusion criteria deviations will also be provided, separately for healthy volunteers and psoriasis patients. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

- There are no planned examination of covariates and subgroups.
- There are no planned adjustments made for multiple centres in this study.
- There are no planned adjustments for multiple comparisons or multiplicity.

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Output | Output |
| Code | Description | Treatment Label | Order |
| A | 0.0003mg/kg GSK2831781 IV single dose | 0.0003mg/kg (ADA-ve) | 2 |
| В | 0.0015mg/kg GSK2831781 IV single dose | 0.0015mg/kg (ADA-ve) | 3 |
| С | 0.0075mg/kg GSK2831781 IV single dose | 0.0075mg/kg (ADA-ve) | 4 |
| D | 0.04mg/kg GSK2831781 IV single dose | 0.04mg/kg (ADA-ve) | 5 |
| Е | 0.15mg/kg GSK2831781 IV single | 0.15mg/kg (ADA-ve) | 6 |
| | dose | 0.15mg/kg (ADA+ve) | 7 |
| | | 0.15mg/kg Combined | 8 |
| F | 0.5mg/kg GSK2831781 IV single dose | 0.5mg/kg | 10 |
| G | 1.5mg/kg GSK2831781 IV single dose | 1.5mg/kg | 11 |
| Н | 5mg/kg GSK2831781 IV single dose | 5mg/kg | 12 |
| P | Placebo IV single dose | Placebo for HV Combined | 1 |
| | | Placebo for PSO | 9 |

#### Notes:

- 1. ADA status as defined at screening
- 2. Combined treatment groups include subjects with ADA-ve and ADA+ve (only for healthy volunteers (HV))

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

Table 2 Baseline Definitions - SAFETY ENDPOINTS

| | Study assessments considered as baseline | | | Baseline used in data display |
|---|---|---|---|---|
| Parameter <sup>1</sup> | Screening Day -1 | | Day 1<br>(pre-<br>dose) | |
| Healthy Volunteers (No DTH) | | | | |
| 12 Lead ECG & Vital Signs | X | Χ | Χ | Day 1 (pre-dose) |
| Lab results | Х | Χ | | Day -1 |
| Cytokine | | | Χ | Day 1 (pre-dose) |
| Psoriasis patients | | | | • |
| Vitals Signs | Х | Х | Χ | Day 1 (pre-dose) |
| 12-Lead ECG | Х | | Χ | Day 1 (pre-dose) |
| Lab results | Х | Х | | Day -1 |
| Cytokines | | | Χ | Day 1 (pre-dose) |

| | Study a | assessments | | | |
|---|---|---|---|---|---|
| Parameter <sup>1</sup> | Day -26 Day -24 dos | | Day 1 (pre-<br>dose) | Baseline used in data display | |
| Healthy Volunteers (DT | H) | | | | |
| Vitals Signs | Χ | X | | X | Day 1 (pre-dose) |
| 12-Lead ECG | Х | | | X | Day 1 (pre-dose) |
| Lab results | Х | | Х | | Day -1 |
| Cytokines | | | | X | Day 1 (pre-dose) |

Table 3 Baseline Definitions – EFFICACY / PHARMACODYNAMIC AND BIOMARKER ENDPOINTS

| Parameter | Visit considered as baseline | | Baseline used for data |
|---|---|---|---|
| | Day -1 | Day 1 (pre-dose) | displays |
| Healthy Volunteers (No DTH) | | | |
| Flow cytometry | | X | Day 1 (pre-dose) |
| G-CSF | | X | Day 1 (pre-dose) |
| sLAG-3 | | X | Day 1 (pre-dose) |
| Blood transcriptomics | | X | Day 1 (pre-dose) |
| Psoriasis patients | | | |
| PBSA | Х | | Day -1 |
| PASI | X | | Day -1 |
| PLSS | X | | Day -1 |
| PGA | X | | Day -1 |
| Flow cytomery | | X | Day 1 (pre-dose) |
| G-CSF | | X | Day 1 (pre-dose) |
| sLAG-3 | | X | Day 1 (pre-dose) |
| Blood transcriptomics | | X | Day 1 (pre-dose) |
| Skin Biopsy (transcriptomics) | X | | Day -1 |

| Parameter | Visit consid | ered as base | line | | Baseline used for data |
|---|---|---|---|---|---|
| | Challenge<br>DTH | Challenge<br>DTH | Challenge<br>DTH Day - | Challenge<br>DTH Day 1 | displays |
| | Day -26 | Day -24 | 1 | (pre-dose) | |
| Healthy Volunteers (D | TH) | | | | |
| Induration [*] | Χ | Χ | | | DTH Day -24 if 2 |
| | | | | | assessments |
| | | | | | DTH Day -26 if only 1 |
| | | | | | assessment |
| | | | | | (see footnote) |
| Flow cytometry | | | | Χ | DTH Day 1 (pre-dose) |
| G-CSF | | | | Х | DTH Day 1 (pre-dose) |
| sLAG-3 | | | | Χ | DTH Day 1 (pre-dose) |
| Blood | | | | Χ | DTH Day 1 (pre-dose) |
| Transcriptomics | | | | | , , , |
| Skin Biopsy - Lag3 | Χ | | | | DTH Day -26 |
| and CD3 | | | | | |
| [*] HV may be re-challer | nged on Day - | 24 if the challe | enge on Day -2 | 26 is not suffici | ent. |

## 6. STUDY POPULATION ANALYSES

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic characteristics, prior and concomitant medications will be based on GSK core data standards.

Screen failures for part A and B will be identified using the cutoff date of 2<sup>nd</sup> June 2016.

Details of the planned displays are presented in Appendix 9.

#### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards.

The details of the planned displays are provided in Appendix 9.

# 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests (at some visits, only liver chemistry and CRP – see e.g. footnote d in T&E for HV (no DTH)), hematology laboratory tests, urinalysis, cytokines and liver function tests will be based on GSK Core Data Standards. In addition, CMV and EBV serology sample will be listed.

Blood samples for viral load monitoring (CMV, EBV, HSV, VZV) taken at baseline and archived will be listed if subsequently analysed (i.e. when a subject demonstrates any clinical symptoms consistent with viral reactivation).

The cytokines are:

- IL-6
- TNF-α
- IL-8
- IFN-γ
- G-CSF

The details of the planned displays are provided in Appendix 9. In tables/figures, if BLQ, LLQ/2 imputed

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results will be based on GSK Core Data Standards, unless otherwise specified. The non-laboratory safety test results include:

- ECGs
- Vital signs

The details of the planned displays are provided in Appendix 9.

### 8. EFFICACY ANALYSES

# 8.1. DTH Induration (only for HV)

# 8.1.1. Endpoint / Variables

- The induration diameter (mm) by challenge site is defined as the average of the 2 skin response test values (vertical and horizontal) at each challenge site.
   A challenge site is defined by skin response (SR) directionality (upper/lower) and SR laterality (left/right). There are 4 categories:
  - Left upper
  - Right upper
  - Left lower
  - Right lower
- 2. The overall induration diameter (mm) is defined as the average of the non-missing induration diameters over the challenge sites.
- 3. The duration of induration is the time (in days) to achieve an overall induration less than 6mm from baseline (see Section 5.2 for baseline definition). It will be calculated as: Date of 1<sup>st</sup> overall induration < 6mm Date of baseline induration assessment + 1. For these subjects who do not achieve an overall induration less than 6mm from the time of the PPD re-challenge post dose, the duration of induration is calculated as time from the PPD re-challenge post dose up to the last available induration measurement +1.

#### 8.1.2. Summary Measure

Induration diameter: absolute and change from baseline for HV (DTH subjects only).

Duration of induration: absolute

Data related to ID PPD challenge will be listed.

### 8.1.3. Population of Interest

The efficacy analyses will be based on the Safety population.

# 8.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.1.4.1. Statistical Methodology Specification

#### **Endpoint**

Change from baseline in induration diameter (mm) (Overall induration diameter only)

#### **Model Specification**

- Mixed models repeated measures (MMRM) model.
- Terms fitted in the MMRM model will include:
  - Fixed categorical covariates: Treatment, day (visit), treatment \* day (visit) interaction
  - Fixed continuous covariates: Baseline (see Section 5.2 for baseline definition)
  - Repeated: Day (visit)
- An unstructured covariance will be used to account for the within-subject correlation. by specifying 'type=UN' on the REPEATED line.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- LSmeans of the CFB will be calculated using the observed margins (OM argument added in the LSmeans function)

#### **Model Checking & Diagnostics**

 In the event that this model fails to converge, alternative correlation structures may be considered.

#### **Model Results Presentation**

Table/Figure of the LS means and 95% CI (by treatment and visit)

#### **Endpoint / Variables**

Duration of induration of at least 6mm (days)

## **Model Specification**

Hasard ratios will be estimated using the Pike estimator.

#### **Model Results Presentation**

- Summary table of the hazard ratios
- No plot

# 8.2. Body Surface Area (only for PsO)

# 8.2.1. Endpoint / Variables

Total body surface area (BSA), in %, measures the area covered with psoriatic plaques.

In the FACE dataset, 4 regional BSA scores (%) are available ((head, upper extremities, trunk, and lower extremities). The total BSA score for each subject at each timepoint is calculated as the sum of the 4 regional BSA scores. If at least one of the 4 regional BSA scores is missing, the total will be set to missing as well.

# 8.2.2. Summary Measure

Absolute BSA scores (4 regional and total), change from baseline and percent change from baseline in BSA scores over time.

#### 8.2.3. Population of Interest

The efficacy analyses will be based on the Safety population.

# 8.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in the section above will be summarised using descriptive statistics, and listed.

# 8.3. PASI-related endpoints (only for PsO)

#### 8.3.1. Endpoint / Variables

Psoriatic lesions will be assessed using the PASI (Psoriasis Assessment Severity Index), single score ranging from 0 (no disease) to 72 (maximal disease). A negative (%) change from baseline in PASI score indicates an improvement.

The PASI score for each subject at each timepoint is derived as follows.

#### Data available (PASI SI dataset):

- Areas of the body: head (1), upper extremities (2), trunk (3), lower extremities (4)
- For each of the 4 areas of the body, the intensity of 3 symptoms is assessed on a 0-4-point rating scale
  - Symptoms: erythema (redness of the skin), induration (thickness) and scaling of the psoriasis

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

• For each of the 4 areas of the body, the percentage area affected by psoriasis is evaluated and expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)

#### **Derivation**

1. Calculation for intensity: the three intensity scores are added up for each of the 4 areas of the body to give 4 subtotals A1, A2, A3, A4.

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

2. Multiply each subtotal (A1, A2, A3, A4) by the body surface area (BSA) represented by that region to give 4 new subtotals (B1, B2, B3, B4).

Note: The BSA will not be calculated using the palm's method as categories above are collected. Fixed weights are used.

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

3. Multiply each subtotal (B1, B2, B3, B4) by the area affected (PASIAREA) for that region to give 4 new subtotals (C1, C2, C3, C4):

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

- 4. Calculate the total PASI score = C1 + C2 + C3 + C4
- 5. If any variable is missing, set PASI score to missing

## 8.3.2. Summary Measure

 Absolute PASI scores, change from baseline and percent change from baseline in PASI scores over time • Proportion of subjects who achieve ≥50% improvement from baseline in PASI score (PASI 50), at each post-baseline visit Proportion of subjects who achieve ≥75% improvement from baseline in PASI score (PASI 75) at each post-baseline visit. If the PASI score is missing, set PASI 50 or 70 to missing.

Note: Day 85 was not assessed for 0.5mg/Kg dosing cohort (cohort 7).

# 8.3.3. Population of Interest

The efficacy analyses will be based on the Safety population.

# 8.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.3.1 will be summarised using descriptive statistics, graphically presented and listed. For the responder endpoints, the exact Binomial 95% CI will be calculated.

#### 8.3.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Change from baseline in PASI scores

#### **Model Specification**

Same MMRM model as for CFB in induration (Section 8.1.4.1)

#### **Model Checking & Diagnostics**

Same approach as in Section 8.1.4.1

#### **Model Results Presentation**

 Table/Figure of the LS means of CFB and 95% CI (by treatment and visit), as well as treatment differences and 95%CI

# 8.4. PLSS-related endpoints (only for PsO)

#### 8.4.1. Endpoint / Variables

The PLSS (Psoriatic Lesion Severity Sum) score for each subject at each timepoint is derived as follows.

#### Data available (CC SI dataset):

For each of the 2 plaques (biopsy or index), the following data will be available:

- The location of the plaque head, face, arm, leg or trunk
- For each plague, the intensity of 3 symptoms is assessed on a 0-4-point rating scale

- Symptoms: induration, erythema, and scaling.
   PLSS total score calculated by the investigator will be in the dataset, but the PLSS score for analysis should be derived from the raw data.
- o 0-4-point rating scale: no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4).

#### Derivation

The PLSS total score for each of the plaques (biopsy and index) is the sum of the scores for the 3 symptoms (induration, erythema, and scaling).

## 8.4.2. Summary Measure

• Absolute PLSS scores, change from baseline and percent change from baseline in PLSS scores over time, for index and biopsy plaques, separately.

## 8.4.3. Population of Interest

The efficacy analyses will be based on the Safety population.

#### 8.4.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.4.1 will be summarised using descriptive statistics, graphically presented and listed.

#### 8.4.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Change from baseline in PLSS scores for the index plaque only

#### **Model Specification**

Same MMRM model as for CFB in induration (Section 8.1.4.1)

#### **Model Checking & Diagnostics**

Same approach as in Section 8.1.4.1

#### **Model Results Presentation**

 Table/Figure of the LS means of CFB and 95% CI (by treatment and visit), as well as treatment differences and 95%CI

# 8.5. PGA-related endpoints (only for PsO)

## 8.5.1. Endpoint / Variables

The Physician Global Assessment (PGA) score for each subject at each timepoint is already in the PGA SI dataset.

A 7-point scoring system will be used to measure the severity of psoriatic lesions over the whole body:



# 8.5.2. Summary Measure

- PGA scores, change from baseline in PGA scores (categories treated as continuous)
- PGA responses (categorical)
- PGA responders defined as subjects achieving PGA 0/1 (clear or almost clear) and at least a 2-point improvement from baseline. This will be performed on subjects with a baseline PGA score of at least 2. Set to missing if baseline PGA is 0 or 1.

## 8.5.3. Population of Interest

The efficacy analyses will be based on the Safety population.

# 8.5.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.5.1 will be summarised using descriptive statistics, graphically presented and listed.

For the responder endpoint, the exact Binomial 95% CI will also be calculated.

#### 9. PHARMACOKINETIC ANALYSES

GUI\_51487 (4.0), effective October 2014, contains the pharmacokinetic methods to be used in non-compartmental analysis (NCA) and reporting of pharmacokinetic studies. This document should be used as a reference.

# 9.1. Drug Concentration Measures

Refer to Section 14.4.3.

#### 9.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin All calculations of non-compartmental parameters will be based on actual

sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable |
| | concentration (C(t)) |
| AUC(0-inf) | Area under the concentration-time curve from time zero and extrapolated to "infinity" |
| Cmax | Maximum observed concentration, |
| tmax | Time to reach Cmax, |
| CL | Clearance |
| t½ | Apparent terminal half-life |
| tlast | Time of last quantifiable concentration |

#### NOTES:

Additional parameters may be included as required.

#### 9.2.1. Population of Interest

The pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 9.2.2. Statistical Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in the section above will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES

## 10.1. IHC parameters

Cells in lesional biopsies are measured by IHC. There are 3 (epidermis thickness is not IHC parameters – separate section) endpoints of interest: LAG3+, CD3+, Ki67 (SI dataset: BIOMARK).

In the dataset, perivascular infiltrates (PVI) cells are also collected:

- HV (DTH): The PVI are used to locate region of interest high power fields (HPFs) for CD3+ and Lag3+ analysis. It is not a biomarker reportable (only listing)
- o PVI is not required for PsO cohorts as regions of interest for HPFs are defined by an alternative approach.

<u>In HV (DTH)</u> LAG3+ and CD3+ were assessed across 3 layers (slices) of the biopsy. A layer represents a section from the lesional skin biopsy tissue. Layers 1-3 represent sections obtained by cutting into the biopsy tissue block at different depths. 10 sections were discarded between each level.

<u>In PsO</u>, LAG3+, CD3+, Ki67 were assessed across 1 layer. The regions of interest (HPFs) for LAG3+ and CD3+ are located in either the epidermis or the superficial dermis. For Ki67, the regions of interest (HPFs) are located in the epidermis only. Epidermal thickness is also only measured in the epidermis.

LAG3+, CD3+ and Ki67 are measured in up to 5 HPFs per layer for HV or epidermis / dermis for PsO. A minimum of 3 HPFs should be present in order for samples to be evaluated.

# 10.1.1. Endpoint / Variables

| Parameter | Endpoint | Derivation | HV<br>(DTH) | PsO |
|---|---|---|---|---|
| LAG3+ | Total number of<br>LAG3+ cells HPFs<br>(A) | For each layer (HV) or epidemis/dermis (PsO) 1. if <b>5 HPFs</b> for <b>all</b> subjects total # of cells (per layer for HV or epidermis/dermis for PsO) = sum of cells in all HPFs (1-5) 2. If <b>3 or 4 HPFs</b> for at least one subject | Y<br>(3<br>layers) | Y<br>(epidermis<br>and<br>dermis) |
| | | Total # of cells of 3/4 HPFs for all subjects = sum of HPFs 1-3, or sum of HPFs 1-4 3. If less than 3 HPFs for some subjects (i.e 0, 1 or 2 HPFs), set to missing for these subjects Note: There is only 1 layer for PsO | | |
| | Total number of LAG3+ cells averaged across skin layers | Sum of (A) as defined above for layers 1, 2 and-3 / 3 layers Note: there will be always 3 layers per subject and timepoint | Υ | N |
| | | Programming notes: 1. Exclude from summary tables/figures if missing (but will be included in listing and individual plots) 2. No LLQ/ULQ for these assays 3. If only some values HPF are missing, it's always in sequential order: e.g. it's not possible to have only HPF2 missing, this should be HPF5 | | |
| CD3+ | Total number of<br>CD3+ cells HPFs<br>(B) | Same derivation as for LAG3+ | Y<br>(3<br>layers) | Y<br>(epidermis<br>and<br>dermis) |
| | Total number of<br>CD3+ cells averaged<br>across skin layers | Same derivation as for LAG3+ | Υ | N |
| | CD3+ (cells/mm²) | (B) as defined above / number of HPFs | N | Υ |

| Parameter | Endpoint | Derivation | HV<br>(DTH) | PsO |
|---|---|---|---|---|
| | | assessed (from 3 to 5 depending on the min number of HPFs available) | | (epidermis<br>and<br>dermis) |
| Perivascular infiltrates (PV) cells | | No derivation | Υ | N |
| Ki67 | Total number of<br>Ki67+ cells HPFs<br>(C) | Same as for as for LAG3+ but only for epidermis | N | Y<br>(epidermis) |
| | Ki67 (cells/mm²) | Same as for CD3+ (cells/mm²) (C) as defined above / number of HPFs assessed (from 3 to 5 depending on the min number of HPFs available) | N | Y<br>(epidermis) |

# 10.1.2. Summary Measure

Absolute, change from baseline and percent change from baseline are of interest for HV and PsO.

Data will be available at baseline and Day 4 (for HV) or Day 29 (for PsO).

## 10.1.3. Population of Interest

The primary pharmacodynamics and biomarker analyses will be based on the Safety population, unless otherwise specified.

#### 10.1.4. Statistical Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 10.1.4.1. Statistical Methodology Specification

## **Endpoint / Variables**

- Change from baseline in
  - LAG3+ (total cells averaged across 3 skin layers for HV and total cells in dermis and epidermis separately for PsO)
  - o CD3+:
    - total cells averaged across 3 skin layers for HV
    - cells per mm<sup>2</sup> in dermis and epidermis separately for PsO
- For epidermis only (PsO), change from baseline in
  - Ki67 (cells/mm)

# **Model Specification**

- Endpoints will be statistically analysed using an ANCOVA model.
- Terms fitted in the model will include: Treatment and baseline

#### **Model Results Presentation**

- Summary table of the LS means and 95% CI for CFB (by treatment)
- [No plot as only 1 post-dose assessment]

# 10.2. Epidermis thickness (only for PsO)

# 10.2.1. Endpoint / Variables

Epidermal thickness is measured by making 35 transect measurements across the entire diameter of the epidermis. The values are in the following SI dataset: MI.

| Parameter | Endpoint | Derivation | HV | PsO |
|---|---|---|---|---|
| | | | (DTH) | |
| Epidermis | Epidermis thickness | Mean of the 35 measurements | N | Υ |
| thickness | (µm) | | | (epidermis) |

## 10.2.2. Summary Measure

Absolute, change from baseline and percent change from baseline are of interest for PsO.

Data will be available at baseline and Day 29 (for PsO).

# 10.2.3. Population of Interest

The primary pharmacodynamics and biomarker analyses will be based on the Safety population, unless otherwise specified.

#### 10.2.4. Statistical Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 10.2.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- For epidermis only (PsO), change from baseline in
  - Epidermis thickness (µm)

## **Model Specification**

- Endpoints will be statistically analysed using an ANCOVA model.
- Terms fitted in the model will include: Treatment and baseline

#### **Model Results Presentation**

- Summary table of the LS means and 95% CI for CFB (by treatment)
- [No plot as only 1 post-dose assessment]

# 10.3. Other PD parameters

## 10.3.1. Endpoint / Variables

The following endpoints are of interest (SI dataset: BIOMARK):

- s-LAG3 parameters no derivation is needed
- Flow cytometry 6 key parameters only described below:

| Marker code | Marker | Type (BITESTCD) | Unit (BISTRESU) |
|-------------|-------------------|------------------|-----------------|
| CDX226 | CD45+ CD3- CD19+ | Concentration | CELLS/UL |
| CDX258 | CD45+ CD3+ CD69+ | Concentration | CELLS/UL |
| CDX444 | CD4+CD45RA+1B4+ | Number of events | COUNT |
| CDX445 | CD4+CD45RA+J11L1+ | Number of events | COUNT |
| CDX446 | CD4+CD45RA-1B4+ | Number of events | COUNT |
| CDX447 | CD4+CD45RA-J11L1+ | Number of events | COUNT |

For 4 of these endpoints (CDX444, CDX445, CDX446, CDX447), the derivation below should be applied (same derivation as for PK analyses):

The count at each time point is the difference: BISTRESN value in the row with BIEXPS = "Stained Sample - T cell markers including J11 and 1B4" - BISTRESN value in the row with BIEXPS = 'LAG3 FMO Control - T cell markers excluding J11 and 1B4'

#### 10.3.2. Summary Measure

- S-LAG3: absolute, change from baseline for <u>total</u> soluble LAG3 concentrations
- Flow cytometry: absolute, change from baseline and <u>percent of baseline</u>, where the percent of baseline is: 100 \* <u>post-dose visit value</u>

  Recelline

## 10.3.3. Population of Interest

The primary pharmacodynamics and biomarker analyses will be based on the Safety population, unless otherwise specified.

#### 10.3.4. Statistical Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.3.1 will be summarised using descriptive statistics, graphically presented and listed.

## 10.4. Transcriptomics (biopsy and blood)

# 10.4.1. Endpoint / Variables

The following endpoints are of interest:

- Blood transcriptomics (HV, PSO):
  - 1. 2 genes: LAG-3 long, LAG-3 short
  - 2. 2 housekeeping genes: POL2RG, POL2RJ
- Biopsy (skin) transcriptomics (PSO only)
  - 1. 18 genes (including the 2 common genes for blood transcriptomics)

| LAG-3 Long | LAG-3 Long Gene mRNA Expression |
|-------------|----------------------------------|
| LAG-3 short | LAG-3 short Gene mRNA Expression |
| IL-17A | IL-17A Gene mRNA Expression |
| IL-17F | IL-17F Gene mRNA Expression |
| IL-22 | IL-22 Gene mRNA Expression |
| IL-23 | IL-23a Gene mRNA Expression |
| IFNg | IFNg Gene mRNA Expression |
| IL-12A | IL-12A Gene mRNA Expression |
| IL-10 | IL-10 Gene mRNA Expression |
| FOXP3 | FOXP3 Gene mRNA Expression |
| S100A12 | S100A12 Gene mRNA Expression |
| Ki67 | Ki67 Gene mRNA Expression |

| K16 | K16 Gene mRNA Expression |
|--------|-----------------------------|
| CD3g | CD3g Gene mRNA Expression |
| TSPAN8 | TSPAN8 Gene mRNA Expression |
| CLDN8 | CLDN8 Gene mRNA Expression |
| CCL27 | CCL27 Gene mRNA Expression |
| CDHR1 | CDHR1 Gene mRNA Expression |

2. 2 housekeeping genes (same as for blood transcriptomics): POL2RG, POL2RJ

## Data available (SI dataset: PF – pharmacogenomics findings):

- Analyte (Collected Specimen Type code): skin or blood
- Gene (Genetic Region of Interest code)
- Type of values (Pharmacogenomics Test code)
  - Cycle times (Ct) 3 per subject
  - Mean of the Cts
  - Delta Ct
  - Delta Delta Ct
  - Fold change

No derivation is needed by S&P as provided by the vendor.

## **10.4.2.** Summary Measure

For all endpoints above:

- Delta delta Ct baseline versus post-baseline visit
- Fold change from baseline to post-baseline visit: always strictly positive (=2^ delta delta Ct)

#### Post-baseline visits:

- HV (DTH and non DTH): Day 2 (Blood only)
- PsO: Day 2 (blood), Day 15 (skin, only cohort 7, removed for cohorts 8 and 9 in amendment 8), Day 29 (skin)

#### 10.4.3. Population of Interest

The transcriptomics analyses will be based on the Safety population, unless otherwise specified.

#### 10.4.4. Statistical Methods

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables will be summarised using descriptive statistics, graphically presented and listed.

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

The PK/PD analyses will be based on the PK population, unless otherwise specified.

The primary goal of this analysis is to characterise the PK/PD relationship of GSK2831781 administered IV in healthy subjects and psoriasis patients. The influence of subject demographics and baseline characteristics will be investigated.

A summary of the planned population PK/PD analyses are outlined below:

- Drug GSK2831781 plasma concentration and corresponding receptor occupancy data will be subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK/PD model.
- To support this analysis a PK/PD dataset will be generated. The details for the dataset specifications are provided in Appendix 7.
- Detailed PK/PD methodology is presented in Appendix 7.

A PK/PD report will be produced by CPMS, and will be included as an appendix to the CSR.

#### 12. IMMUNOGENICITY ANALYSES

The immunogenicity analyses will be based on the Safety population, unless otherwise specified.

Information from the screening assay contributes to the number at risk for the calculation of % positive. The calculation of 'n' is displayed in the diagram below as a guide.



There are no planned statistical analyses.

Details of the planned displays are provided in Appendix 9 and will be based on GSK data standards and statistical principles.

# 13. BAYESIAN ANALYSES (PART B)

To aid decision making, the following posterior probabilities, will be evaluated:

#### For **PASI/PLSS**:

- Difference of interest = Difference (active placebo) in % CFB,
- Probabilities of interest

P(difference < 0)  $P(difference \le 10\%)$   $P(difference \le 20\%)$   $P(difference \le 30\%)$  $P(difference \le 40\%)$ 

### For **total LAG3 cells** for the epidermis and dermis:

- Difference of interest = Difference (active placebo) in % CFB
- Probabilities of interest

P(difference < 0) $P(difference \le 30\%)$ 

#### For Ki67 and epidermis thickness:

- Difference of interest = Difference (active placebo) in CFB
- Probabilities of interest

P(difference < 0)

The active and placebo treatment groups mentioned above are defined as follows:

- Subjects in the active group are defined as psoriasis patients that received the doses 1.5mg/kg and 5mg/kg (pooled cohorts 8 and 9). In total, 12 subjects are on active.
- Subjects in the placebo group are defined as psoriasis patients that received placebo in cohorts 7-9. In total, 9 subjects are on placebo.

The propobabilities described above may also be calculated for each dose (i.e. 1.5mg/kg versus placebo and 5mg/kg versus placebo).

For PASI and PLSS, the change from baseline to lowest non-missing post-baseline response will be derived for each subject, considering all their available assessments out to day 85. The Bayesian analyses will be conducted for these derived endpoints to provide an overall summary, as oppose to a distinct assessment at each timepoint. For the other endpoints changes from baseline to day 29 will be assessed.

Changes from baseline in each parameter will be analysed using a linear regression, including treatment (active and control as defined above) and baseline score:

 $Y_i \sim \text{Normal}(\mu_i, \text{precision} = \tau)$  $\mu_i = \beta_0 + \beta_1 Base_i + \beta_2 Treatment_i$  Where  $Y_i$  is the observed change from baseline response for each subject as defined above.

Non-informative conjugate prior distributions are assigned to the unknown parameters:

- Intercept and slope coefficients:  $\beta_0$ ,  $\beta_1$ ,  $\beta_2 \sim \text{Normal}(0, \text{precision} = 10^{-3})$ Sensitivity analysis with precion=0.1
- Between-subject precision (1/variance):  $\tau \sim$  Gamma (shape = 0.001, rate = 0.001), i.e.  $E(\tau) = 1$

One MCMC chain will be run. At least 10 000 iterations will be used for the burn-in period as well as for the inference. The number of iterations may be increased to ensure that the ratio MCSE/SD for all the parameters in the model is  $\leq 0.01$ .

Visual inspection of MCMC output (including, but not limited to, trace and autocorrelation plots) will be used to assess the convergence.

The posteriror distribution of the difference in % CFB will be generated as  $\beta_2$  /  $mean\_Base$ . The later is modelled as a normal distribution and assumed that there is no treatment difference for baseline values before treatment:  $Base_i \sim Normal(mean\_Base,$  precision =  $\tau\_Base$ ). Non-informative conjugate prior distributions are assigned to the unknown parameters:

- mean Base  $\sim$  Normal(0, precision =  $10^{-3}$ )
- Between-subject precision (1/variance):  $\tau$ \_Base ~ Gamma (shape = 0.001, rate = 0.001), i.e.  $E(\tau) = 1$

The posterior probabilities that the difference in %CFB or CFB is above a pre-defined threshold will be calculated based on the above posterior distributions.

Results will be displayed in a table, with the number of subjects in each group, active and control.

# 14. APPENDICES

# 14.1. Appendix 1: Protocol Defined Schedule of Events

# 14.1.1. Healthy volunteers (no DTH)

| Protocol Activity | Base-<br>line | | In Clinic Period | | | | | | | | | | Out Patient Visits | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | ay 1 | | | Day 2 | Day 3 | Day 4 | Day 8 | | | | | | | | | | |
| | Day -1 | Pre-<br>dose | 0 hour | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post-<br>infusion<br>start | | | 24 hour<br>post-<br>infusion<br>start | | | 168<br>hour<br>post-<br>infusion<br>start | Day<br>11 | Day<br>15 | Day<br>18 | Day<br>22 | Day<br>25ª | Day<br>29 <sup>k</sup> | Day<br>43 | Day<br>571 | Day<br>85 | Day<br>121 |
| Window | | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±3d |
| Admission to the<br>unit | X | | | | | | | | | | | | | | | | | | | | |
| Discharge from<br>the unit | | | | | | | | | | Х | | | | | | | | | | | |
| Brief physical | Χ | | | | | | | | | | | | | | | | | | | | |
| Urine Drug and<br>Alcohol Screen | Х | | | | | | | | | | | | | | | | | | | | |
| Administer IV<br>Dose (2 hour<br>infusion) | | | <b>4</b> | <b>&gt;</b> i | | | | | | | | | | | | | | | | | |
| Safety Assessme | ents | | | | | - | | | | - | | | | | | | | | | | $\neg$ |
| Vital Signs | Χ | X | | X | X | X | X | X | Х | X | X | | Χ | | Χ | | X | Χ | Χ | X | Χ |
| 12 - Lead<br>ECG | Χi | Χ | <b>◄</b> | ▶□ | | Х | | | | Х | | | | | | | | | | | |
| Concomitant<br>Medications | <b>◄</b> | | | | | | | | | | | | | | | | | | | | |
| Adverse<br>Events<br>Assessment<br>/ SAE'sc | <b>4</b> | | | | | | | | | | | | | | | | | | | | |
| Laboratory Asses | | s | | | | | | | | | | | | | | | | | | | |
| Haematology | X | | | | | X | X | | | X | X | X | X | X | X | X | X | Х | Χ | X | X |
| Chemistry | X | | | | | Χq | Χα | | | X | X | | X | | Х | | Χ | Х | Χ | X | X |
| Urinalysis | X | | | | | X | X | | | X | X | | X | | X | | X | Х | Χ | X | X |

| Protocol Activity | Base-<br>line | | In Clinic Period | | | | | | | | | | Out Patient Visits | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | ay 1 | | | Day 2 | Day 3 | Day 4 | Day 8 | | | | | | | | | | |
| | Day -1 | Pre-<br>dose | 0 hour | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post-<br>infusion<br>start | 6 hour<br>post-<br>infusion<br>start | 12 hour<br>post-<br>infusion<br>start | post- | post- | 72 hour<br>post-<br>infusion<br>start | 168<br>hour<br>post-<br>infusion<br>start | Day<br>11 | Day<br>15 | Day<br>18 | Day<br>22 | Day<br>25ª | Day<br>29k | Day<br>43 | Day<br>571 | Day<br>85 | Day<br>121 |
| Window | | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±3d |
| CMV and<br>EBV<br>serology<br>sample | х | | | | | | | | | | | | | | | | | | | | |
| Viral load<br>sample<br>(CMV, EBV,<br>HSV, VZV) <sup>e</sup> | x | | | | | | | | | | | | | | | | | | | | |
| PK Samplef | | | | | | <b>4</b> | | | | | | | | | <b>•</b> | | | | | | |
| Immunogenicity<br>Sample | | Х | | | | | | | | | Х | | | | | | Х | | | х | |
| Immune Cell<br>Phenotypings | | Х | | | | Х | | Х | | Х | Х | | Х | | | | Х | | Х | х | х |
| CD16 and LAG-3<br>Receptor<br>occupancy | | Х | | | | Х | | Х | | Х | Х | | х | | | | х | | х | Х | X |
| Cytokine Sample | | Χ | | | | Х | Х | Х | Х | | | | | | | | | | | | |
| G-CSF Sample | | Χ | | | | Х | | Х | | Х | Х | | Χ | | | | Х | Х | Χ | Х | Х |
| sLAG-3 Sample | | Χ | | | | X | | X | | X | X | | Х | | | | Х | Х | Χ | Х | Х |
| Blood<br>Transcriptomics<br>Sample | | X | | | | | | х | | | | | | | | | | | | | |
| Ex Vivo<br>Antigen/Cytokine<br>Stimulation Test | | X | | | | | | Х | | | | | | | | | | | | | |

| Protocol Activity | Base-<br>line | | | | In | Out Patient Visits | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | ay 1 | | Day 2 | Day 3 | Day 4 | Day 8 | | | | | | | | | | |
| | Day -1 | Pre-<br>dose | Pre- 0 hour post- post- post- post- | | | | | post- | post- | nour<br>nost- | Day<br>11 | Day<br>15 | Day<br>18 | Day<br>22 | Day<br>25ª | Day<br>29k | Day<br>43 | Day<br>571 | Day<br>85 | Day<br>121 |
| Window | | | | | | Ĺ . | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±3d |
| In vitro LAG-3+<br>activity | | Х | | Х | | | | | | Х | | | | | | | | | | |
| PGx Sample | Χħ | | | | | | | | | | | | | | | | | | | $\Box$ |

- x oampie X:

  Cohort 0.0003mg/kg last out patient visit will be on Day 25.

  Continuous 2-lead ECG during infusion. Only significant abnormalities during this time will be databased.

  A targeted physical examination may take place if guided by AE reporting relating to Section 6.3.4, Section 6.3.5 and Section 6.3.6..

  Liver Chemistry and CRP only

- Viral load sample for storage as baseline. If symptoms suggestive of viral infection develop then a sample will be taken and analysed with the baseline sample (See Section 6.3).
   See Pharmacokinetic time and events table for dose specific timepoints.
   Additional blood samples may be taken during the study if subject develops infection in order to measure LAG-3+ cells or other parameters as may be clinically or immunologically
- Pharmacogenetics sample can be taken any time after consent is signed.
  To calculate the correct dose, weight must be measured on Day -1 or Day 1 pre-dose.
  Triplicate. Only required if screening ECG not within 35 days of Day 1.
  Cohort 0.0015mg/kg last out patient visit will be on Day 29.
  Cohort 0.0075mg/kg last out patient visit will be on Day 57.
# 14.1.2. Healthy volunteers (DTH subjects)

| Protocol Activity | | st<br>lenge | | | | | In C | linic Per | iod | | | | | | | | Out P | atient | Visits | , | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Day<br>28 | | | Day | 29 (Day 1 | 1) | | Day 30<br>(Day 2<br>post-<br>dose) | Day 31<br>(Day 3<br>post-<br>dose) | Day 32<br>(Day 4<br>post-<br>dose) | | | | | | | | | | | |
| | Day<br>1 | Day 3 | Day<br>28 | Pre-<br>dose | 0<br>hour | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post-<br>infusion<br>start | post- | 12 hour<br>post-<br>infusion<br>start | post- | hours | 72 hour<br>post-<br>infusion<br>start | (Day<br>8<br>post- | | 15<br>post- | 18<br>post- | 22<br>post- | 25<br>post- | 29<br>post- | 43<br>post- | Day<br>85<br>(Day<br>57<br>post-<br>dose) | 85<br>post- | |
| Window | | | ±3d | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±3d |
| Admission to the<br>unit | | | Х | | | | | | | | | | | | | | | | | | | | |
| Discharge from<br>the unit | | | | | | | | | | | | X | | | | | | | | | | | |
| Brief Physical | Х | | Х | | | | | | | | | | | | | | | | | | | | |
| Urine Drug and<br>Alcohol Screen | Χ | | | | | | | | | | | | | | | | | | | | | | |
| Administer IV<br>Dose (2 hour<br>infusion) | | | | | <b>4</b> | n | | | | | | | | | | | | | | | | | |
| Safety Assessme | nts | | | | | | | | | | | | | | | | | | | | | | |
| Vital Signs | Χ | X | | Χ | | X | X | X | X | X | X | X | X | | Χ | | Χ | | X | X | X | Χ | X |
| 12 - Lead<br>ECG | Χa | | | Х | <b>⋖</b> | b | | Х | | | | X | | | | | | | | | | | |
| Concomitant<br>Medications | <b>∢</b> | | | | | | | | | | | | | | | | | | | | | | |
| Adverse<br>Events<br>Assessment<br>/ SAE'sc | <b>4</b> | | | | | | | | | | | | | | | | | | | | | | |

| Protocol Activity | | st<br>lenge | | | | | In C | linic Per | iod | | | | | | | | Out P | atient | Visits | , | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Day<br>28 | | | Day | 29 (Day 1 | 1) | | Day 30<br>(Day 2<br>post-<br>dose) | | Day 32<br>(Day 4<br>post-<br>dose) | | | | | | | | | | | |
| | Day<br>1 | Day 3 | Day<br>28 | | 0<br>hour | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post-<br>infusion<br>start | post- | 12 hour<br>post-<br>infusion<br>start | post- | 48<br>hours<br>post-<br>infusion<br>start | 72 hour<br>post-<br>infusion<br>start | 8<br>post- | 11<br>post- | 15<br>post- | | | | | 43<br>post- | Day<br>85<br>(Day<br>57<br>post-<br>dose) | | 149<br>(Day<br>121<br>post- |
| Window | | | ±3d | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±3d |
| Efficacy Assessn | nents | • | | • | • | | | | | | | | • | • | | | _ | | • | _ | | | • |
| Visual Arm<br>Inspection | Χα | | | | | | | | | Χe | | | | | | | | | | | | | |
| ID PPD<br>Challenge | Χ <sup>f</sup> | | | | | | | | | Хf | | | | | | | | | | | | | |
| Bleb/ILH<br>Assessment | Χe | | | | | | | | | Χe | | | | | | | | | | | | | |
| Ball Point<br>Pen<br>Technique | | Х | | | | | | | | | | Х | х | | Х | | Х | | | | | | |
| Skin Biopsy | | Χg | | | | | | | | | | Χg | | | | | | | | | | | |

| | _ | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activity | | st<br>lenge | | | | | In C | linic Per | iod | | | | | | | | Out F | atient | Visits | • | | | |
| | | | Day<br>28 | | | Day | 29 (Day 1 | 1) | | Day 30<br>(Day 2<br>post-<br>dose) | Day 31<br>(Day 3<br>post-<br>dose) | Day 32<br>(Day 4<br>post-<br>dose) | | | | | | | | | | | |
| | Day<br>1 | Day 3 | Day<br>28 | Pre-<br>dose | 0<br>hour | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post-<br>infusion<br>start | post- | 12 hour<br>post-<br>infusion<br>start | post- | 48<br>hours<br>post-<br>infusion<br>start | start | (Day<br>8<br>post- | | | | | | | | Day<br>85<br>(Day<br>57<br>post-<br>dose) | | |
| Window | | | ±3d | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±3d |
| Laboratory Asses | ssmei | nts | | | | | | | | | | | | | | | | | | | | | |
| Haematology | Χh | | X | | | | | X | X | | | X | X | Х | Х | Х | X | X | X | Χ | Х | Х | X |
| Chemistry | Χh | | Х | | | | | Χi | Χi | | | X | Х | | Х | | Χ | | Χ | Х | Χ | Χ | Χ |
| Urinalysis | Χħ | | Х | | | | | X | Х | | | X | Χ | | Χ | | Х | | Х | Χ | Х | Х | Х |
| CMV and<br>EBV<br>serology<br>sample | | | х | | | | | | | | | | | | | | | | | | | | |
| Viral load<br>sample<br>(CMV, EBV,<br>HSV, VZV)i | | | х | | | | | | | | | | | | | | | | | | | | |
| Immunogenicity<br>Sample | | | | X | | | | | | | | | Х | | | | | | Х | | | Х | |
| PK Sample <sup>k</sup> | | | | | ◀ | | | | | | | | | | | | | | | | ▶ | | |
| Immune Cell<br>Phenotyping | | | | Х | | | | Х | | Х | | Χ | Χ | | X | | | | Х | | X | Χ | X |
| CD16 and LAG-3<br>Receptor<br>occupancy | | | | х | | | | Х | | Х | | Х | Х | | Х | | | | Х | | Х | Х | Х |
| Cytokine Sample | | | | X | | | | X | X | X | X | | | | | | | | | | | | |
| G-CSF Sample | | | | Χ | | | | X | | X | | X | Χ | | Χ | | | | Χ | Χ | Χ | Χ | Χ |

| Protocol Activity | 1<br>Chal | st<br>lenge | | | | | In C | linic Per | iod | | | | | | | Out P | atient | Visits | , | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Day<br>28 | | | Day | 29 (Day 1 | 1) | | Day 30<br>(Day 2<br>post-<br>dose) | Day 31<br>(Day 3<br>post-<br>dose) | Day 32<br>(Day 4<br>post-<br>dose) | | | | | | | | | | |
| | Day<br>1 | Day 3 | Day<br>28 | Pre-<br>dose | 0<br>hour | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post-<br>infusion<br>start | post- | post- | 24 hour<br>post-<br>infusion<br>start | 48<br>hours<br>post-<br>infusion<br>start | 72 hour<br>post-<br>infusion<br>start | (Day<br>8<br>post- | | 15<br>post- | 22<br>post- | | 29<br>post- | | Day<br>85<br>(Day<br>57<br>post-<br>dose) | | |
| Window | | | ±3d | | | | | | | | | | _ | ±1d | _ | _ | _ | _ | | ±2d | | ±3d |
| sLAG-3 Sample | | | | Χ | | | | X | | Х | | Х | Χ | | Χ | | | Χ | Х | Х | Χ | Χ |
| Blood<br>Transcriptomics<br>Sample | | | | X | | | | | | Х | | | | | | | | | | | | |
| Ex vivo<br>antigen/cytokine<br>stimulation | | | | х | | | | | | Х | | | | | | | | | | | | |
| In vitro LAG-3+<br>activity | | | | X | | Х | | | | | | | X | | | | | | | | | |
| PGx Sample | Χm | | | | | | | | | | | | | | | | | | | | | |

- Triplicate. Only required if screening ECG not within 35 days of Day 1.
   Continuous 2-lead ECG during infusion. Only significant abnormalities during this time will be databased.
- A targeted physical examination may take place if guided by AE reporting relating to Section 6.3.4, Section 6.3.5 and Section 6.3.6.
- d. Must be performed before ID PPD Challenge
- Bleb is assessed 5 minutes after ID injection and the immediate local hypersensitivity assessment 15-30 minutes after ID injection. See Section 5.10.1 for details.
- g. Only biopsy from one of the PPD sites preferably from the subjects non-dominant arm.
- h. If safety labs have been taken ≤7 days prior to challenge then these safety labs are not required. These samples can be taken on Day 1 or Day -1.
- Liver Chemistry and CRP only
- Viral load sample for storage as baseline. If symptoms suggestive of viral infection develop then a sample will be taken and analysed with the baseline sample (See Section
- 6.3).
  See Pharmacokinetic time and events table for dose specific timepoints.
  Additional blood samples may be taken during the study if subject develops infection in order to measure LAG-3+ cells or other parameters as may be clinically or
- m. Pharmacogenetics sample can be taken any time after consent is signed.
- To calculate the correct dose, weight must be measured on Day 28 or Day 29 pre-dose.

# 14.1.3. Psoriasis patients

| Protocol Activity | Base-<br>line | | | | ı | n Clinic | Period | | | | | | | | 0 | ut Pati | ent Vi | isits <sup> </sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Day 1 | | | Day 2 | Day 3 | Day 4 | Day 8 | | | | | | | | | | | | П |
| | Day - | | | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post-<br>infusion<br>start | post- | post- | 24 hour<br>post-<br>infusion<br>start | post- | post- | | | Day<br>15 | Day<br>18 | Day<br>22 | Day<br>25 | Day<br>29 | Day<br>36 n | Day<br>43 | Day<br>57 | Day<br>71 n | Day<br>85 | Day<br>121 |
| Window | | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±2d | ±3d |
| Admission to the<br>unit | Х | | | | | | | | | | | | | | | | | | | | | | |
| Discharge from<br>the unit | | | | | | | | | | Х | | | | | | | | | | | | | |
| Reassess 2 target<br>lesions for<br>suitability | Х | | | | | | | | | | | | | | | | | | | | | | |
| Brief physical | X | | | | | | | | | | | | | | | | | | | | | | |
| Urine Drug and<br>Alcohol Screen | X | | | | | | | | | | | | | | | | | | | | | | |
| Administer IV<br>Dose (2 hour<br>infusion) | | | 4 | <b>→</b> j | | | | | | | | | | | | | | | | | | | |
| Safety Assessme | nts | - | - | | | | | - | | - | | - | - | - | | | - | - | | | | | _ |
| Vital Signs | Χ | Χ | | X | X | Х | X | X | X | X | X | | Χ | | Х | | Χ | | Х | Х | | Χ | Х |
| 12 - Lead ECG | Χk | Х | 4 | <b>&gt;</b> a | | X | | | | X | | | | | | | | | | | | | |
| Concomitant<br>Medications | | | | <b>∢</b> | | | | | | | | | | | | | | | | | | | |
| Adverse Events /<br>SAEs ¤ | | | | <b>∢</b> | | | | | | | | | | | | | | | | | | , | |

| Protocol Activity | Base- | | | n Clinic | Period | | | | | | | | Oı | ut Pati | ent Vi | sits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Day 1 | | | Day 2 | Day 3 | Day 4 | Day 8 | | | | | | | | | | | | |
| | Day - | 2 hour<br>post-<br>infusion<br>start | 4 hour<br>post- | post- | 12 hour<br>post-<br>infusion<br>start | 24 hour<br>post- | 48 hour<br>post- | 72 hour<br>post- | 168<br>post- | | Day<br>15 | Day<br>18 | Day<br>22 | Day<br>25 | Day<br>29 | Day<br>36 n | Day<br>43 | Day<br>57 | Day<br>71 n | Day<br>85 | Day<br>121 |
| Window | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±2d | ±3d |
| Efficacy Assessn | nents | - | - | - | - | - | | | | • | • | | | | | | | | - | | • |
| Psoriatic<br>Body<br>Surface Area | X | | | | | | | | | | Х | | | | X | | X | | | X | X |
| Psoriasis<br>Area<br>Severity<br>Index | x | | | | | | | | | | х | | | | x | | X | | | x | X |
| Psoriatic<br>Lesion<br>Severity<br>Score | Χ¢ | | | | | | | | | | Χ¢ | | | | Χ¢ | | Χď | | | Χq | Χď |
| Phys. Global<br>Assessment<br>Scale | X | | | | | | | | | | х | | | | X | | X | | | х | x |
| Skin Biopsy | Х | | | | | | | | | | | | | | Х | | | | | | |
| Photograph<br>of index<br>lesion | X | | | | | | | | | | Х | | | | х | | X | | | Х | x |
| Photograph<br>of biopsy<br>lesion e | X | | | | | | | | | | | | | | х | | | | | | |

| Protocol Activity | Base-<br>line | | | | ı | n Clinic | Period | | | | | | | | Oı | ıt Pati | ent V | sits <sup> </sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Day 1 | | | Day 2 | Day 3 | Day 4 | Day 8 | | | | | | | | | | | | |
| | | | | 2 hour | 4 hour | 6 hour | 12 hour | 24 hour | 48 hour | 72 hour | 168 | | | | | | | | | | | | |
| | Day - | Pre- | 0 | post- | post- | post- | post- | post- | post- | post- | post- | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day |
| | 1 | dose | hour | infusion | infusion | infusion | infusion | infusion | infusion | infusion | infusion | 11 | 15 | 18 | 22 | 25 | 29 | 36 n | 43 | 57 | 71 n | 85 | 121 |
| | | | | start | start | start | start | start | start | start | start | | | | | | | | | | | | |
| Window | | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±2d | ±3d |
| Laboratory Asse | ssmen | ts | | | | | | | | | | _ | | | | | | | _ | | | | _ |
| Haematology | X٥ | | | | | X | Χo | | | Χo | Χo | Χ | X | Х | Х | Х | Χ | | X | Χ | | Χ | X |
| Chemistry | Χ | | | | | Χf | Χf | | | Х | Х | | Х | | Х | | Х | | Χ | Χ | | Х | Х |
| Urinalysis | Х | | | | | Х | Х | | | Х | Х | | Х | | Х | | Х | | Х | Х | | Х | Х |
| Urine | | | | | | | | | | | | | | | | | | | | | | | $\Box$ |
| Pregnancy<br>Test (FRP) | Х | | | | | | | | | | | | | | | | X | | | X | | Χ | X |
| CMV and<br>EBV<br>serology<br>sample | х | | | | | | | | | | | | | | | | | | | | | | |
| Viral load<br>sample<br>(CMV, EBV,<br>HSV, VZV) <sup>9</sup> | х | | | | | | | | | | | | | | | | | | | | | | |
| Immunogenicity<br>Sample | | Χ | | | | | | | | | Χ | | | | | | Χ | | | | | χ | |
| PK Sample h | | | | ◀ | | | | | | | | | | | | | | | | | | | |
| Immune Cell<br>Phenotyping i<br>(Flow) | | х | | | | Х | | х | | Х | Х | | х | | | | х | | х | X | | х | X |
| Immune Cell<br>Phenotyping <sup>m</sup><br>(Chip) | | х | | 4- | | | | | | | | m | | | | | | | | | | | |
| CD16 and LAG-3<br>Receptor<br>occupancy | | Х | | | | X | | X | | Х | Х | | X | | | | Х | | Х | X | | Х | x |

| Protocol Activity | Base-<br>line | | | | ı | n Clinic | Period | | | | | | | | 0 | ut Pati | ient Vi | sits ! | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Day 1 | | | Day 2 | Day 3 | Day 4 | Day 8 | | | | | | | | | | | | |
| | | | | 2 hour | 4 hour | 6 hour | 12 hour | 24 hour | 48 hour | 72 hour | 168 | | | | | | | | | | | | |
| | Day - | | | post- | post- | post- | post- | post- | post- | post- | post- | | | Day | | | | | | | Day | | |
| | 1 | dose | hour | infusion | infusion | infusion | infusion | infusion | infusion | infusion | infusion | 11 | 15 | 18 | 22 | 25 | 29 | 36 n | 43 | 57 | 71 n | 85 | 121 |
| | | | | start | start | start | start | start | start | start | start | | | | | | | | | | | | |
| Window | | | | | | | | | | | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±1d | ±2d | ±2d | ±2d | ±2d | ±3d |
| Cytokine Sample | | Χ | | | | Х | X | Х | X | | | | | | | | | | | | | | |
| G-CSF Sample | | Х | | | | Х | | X | | X | X | | Х | | | | Х | | Х | Х | | Χ | Х |
| sLAG-3 Sample | | Χ | | | | X | | X | | Х | X | | Χ | | | | Χ | | Χ | Χ | | Χ | Х |
| Blood | | | | | | | | | | | | | | | | | | | | | | | |
| Transcriptomics | | X | | | | | | X | | | | | | | | | | | | | | | |
| Sample | | | | | | | | | | | | | | | | | | | | | | | |
| PGx Sample | Х | | | | | | | | | | | | | | | | | | | | | | |

- Continuous 2-lead ECG during infusion. Only significant abnormalities during this time will be databased.
- A targeted physical examination may take place if guided by AE reporting relating to Section 6.3.4, Section 6.3.5 and Section 6.3.6.
- PLSS will be recorded for the index lesion and the biopsy lesion (prior to the biopsy being performed).
- c. d. Index lesion only.
- Photographs of the biopsy lesion will be taken before the skin biopsy.
- Liver Chemistry and CRP only
- Viral load sample for storage as baseline. If symptoms suggestive of viral infection develop then a sample will be taken and analysed with the baseline sample (See Section 6.3).
- See Pharmacokinetic time and events table for dose specific timepoints.
- Additional blood samples may be taken during the study if e.g. subject develops infection (measure LAG-3+ cells), hypersensitivity reactions (serum tryptase), signs/symptoms suggestive of viral reaction, or other parameters as may be clinically or immunologically indicated (See Section 6.3).
- To calculate the correct dose, weight must be measured on Day -1 or Day 1 pre-dose. Triplicate. Only required if screening ECG not within 35 days of Day 1.
- Investigator/designee should remind subjects to comply with contraception requirements on an ~ monthly basis until Follow-Up (either at study visits or by telephone call).
- Immune Phenotyping (Chip) Cohort 7: at Baseline, 6 hours post-start of infusion, Day 8 and 15. Cohorts 8 and 9: at Baseline, 6 hours post start of infusion, Day 43 and 85.
- Additional visit introduced at Day 36 (Cohort 8 only) and Day 71 (Cohort 9 only).

  Samples taken for haematology at Day -1, 12 hours, 72 hours and 168 hours are to include analysis for CD3, CD4 and CD8 lymphocyte subsets.

# 14.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

### 14.2.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior, and up to the last scheduled visit attended (follow-up or combined FU/surveillance) |
| Off-treatment | Medication started between the last scheduled visit and the surveillance visit will be included in the listing, and flagged. |
| | 5 for handling of missing and partial dates for concomitant medication. Use the rules in itant medication date is completely missing. |

### 14.2.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Prior | Any starting date before 1st dose |
| Treatment<br>Emergent | Any starting date between 1st dose and last scheduled visit (follow-up or combined FU/surveillance) |
| Off treatment | AE occurring between the last scheduled visit and the surveillance visit will be included in the listing, and flagged. |
| Refer to Appendix completely missing. | 5 for handling of missing and partial dates for AE. Use the rules in this table if date is |

#### 14.3. Appendix 3: A&R Data sets

#### 14.3.1. Subject-Level Variables

#### 14.3.1.1. ADA Status

ADASTACD/ADASTAT should be included in POP, AE plus any other data sets with outputs split by ADA status.

- If a subject has one "positive" record for the confirmatory assayin IMGEN (IGSCATCD=2 and IGORRSCD=1) at <u>screening</u> then set to positive (ADASTATCD=1 / ADASTAT="ADA Positive")
- Otherwise set to negative (ADASTATCD=2 / ADASTAT="ADA Negative")

#### 14.3.1.2. Treatment

TRTCD/TRTGRP should be completed as specified in RAP Section 5.1.

Complete as follows:

- 1. Merge DM data sets RAND and RANDALL by RANDNUM to get the PTRTGRP and SCHEDNUM/SCHEDTX for each SUBJID.
- 2. TRTCD/TRTGRP are then completed from PTRTGRP and SCHEDNUM as described below.
- 3. Check the ADA status (IMGEN screening data) of all subjects compared with the treatment group assignment.
- 4. Unrandomised subjects (i.e. subjects with no RANDNUM) will have TRTCD/TRTGRP missing.
- 5. The actual treatment variables ATRTCD/ATRTGRP should just be copied from TRTCD/TRTGRP unless any subject is known to have taken the wrong treatment. In addition, ATRTCD/ATRTGRP can be set to 888/"No Treatment" for untreated subjects as in the SPOTFIRE version of POP.

# 14.4. Appendix 4: Data Display Standards & Handling Conventions

### 14.4.1. Reporting Process

| Software | |
|---|---|
| The currently supply | ported versions of SAS software will be used. |
| Reporting Area | . • |
| HARP Server | . • |
| HARP Compound | |
| <b>Analysis Datasets</b> | |
| Analysis datasets | Analysis datasets will be created according to Legacy GSK A&R dataset standards. |
| Generation of RTF Fi | Generation of RTF Files |
| RTF files will be get a second control of the second control | enerated for Interim 2 and SAC. |

#### 14.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
- Under Supporting Documentation > Component > Statistical Displays
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| <b>Unscheduled Visits</b> | |
|---|---|
| <ul> <li>Unscheduled visit</li> </ul> | s will not be included in by-visit summary tables and figures. |
| <ul> <li>Unscheduled visit</li> </ul> | s will be considered when deriving maximum/worse post-baseline values. |
| All unscheduled v | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | |
| Categorical Data | · |
| <b>Graphical Displays</b> | |
| Refer to IDSL Sta | tistical Principals 7.01 to 7.13. |
| Laboratory Paramete | ers |
| detectable level re<br>character value st | If a laboratory value which is expected to have a numeric value for summary purposes, has a non-<br>detectable level reported in the database, where the numeric value is missing, but typically a<br>character value starting with ' <x' '="" or="">x' (or indicated as less than x or greater than x in the comment<br/>field) is present, the number of significant digits in the observed values will be used to determine how</x'> |

Example 1: 2 Decimal Places= '< x ' becomes x – 0.01</li>

much to add or subtract in order to impute the corresponding numeric value.

- O Example 2: 1 Decimal Place= '> x' becomes x + 0.1
- Example 3: 0 Decimal Places= '< x' becomes x 1

### 14.4.3. Reporting Standards for Pharmacokinetic

| Concentration Data | |
|---|---|
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Pharmacokinetic Para | ameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and [between and or within] geometric coefficient of variation (CVb/w (%)) will be reported. [1] $CV_b$ (%) = $\sqrt{\exp(SD^2) - 1} * 100$ (SD = SD of log transformed data) [2] $CV_w$ (%) = $\sqrt{\exp(MSE) - 1} * 100$ (MSE = mean square error from mixed effect model of loge-transformed data). |
| Parameters Not<br>Being Log<br>Transformed | tmax, tlast |

# 14.5. Appendix 5: Reporting Standards for Missing Data

# 14.5.1. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 14.5.1.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered as treatment-emergent.</li> <li>Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 14.6. Appendix 6: Values of Potential Clinical Importance

# 14.6.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | a/I | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| - | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | $\geq 2x$ ULN ALT |

#### 14.6.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase in Baseline in QTc | msec | | >60 |

The following categories will be used for summarising by:

- the maximum QTc values post-baseline relative to baseline
- the maximum increase in QTc values post-baseline relative to baseline

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | < 450 | |
| Absolute QTcB and QTcF Interval | msec | ≥ 450 | ≤ 479 |
| | | ≥ 480 | ≤ 500 |
| | | > 500 | |
| 0, , , , , , | msec | < 30 | |
| Change from baseline in QTcB and QTcF | | ≥ 30 | ≤ 60 |
| WICD allu WICF | | > 60 | |

### 14.6.3. Vital Signs

| Vital Sign Parameter | Units Clinical Concern Range | | cern Range |
|--------------------------|------------------------------|-------|------------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

### 14.7. Appendix 7: Pharmacokinetic/Pharmacodynamic Analyses

All non-linear mixed effects modelling will be performed using NONMEM (ICON Solutions), PsN (Perl Speaks NONMEM) and Pirana (Pirana Software & Consulting BV 2016).

R (The R Foundation for Statistical Computing) will be used for exploratory graphical analysis, graphical model diagnostics and, if needed, modifications of the dataset.

The analysis will be performed by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline in the GSK modelling environment MAP (Model-based Analyses Platform) using the currently supported versions of all software packages.

#### 14.7.1. Pharmacokinetic / Pharmacodynamic Dataset Specification

The merging of aLAG3, regiment, biomarker and demographic data together with the creation of the NONMEM-specific dataset will be performed by, or under the direct auspices of, Clinical Statistics (Programmer), GlaxoSmithKline.

This dataset programming will be conducted in a HARP environment using the currently supported version of SAS.

### 14.7.2. Pharmacokinetic / Pharmacodynamic Methodology

An exploratory graphical analysis of the data will be performed by generating the plots as presented in Appendix 9.

Model development will be data driven.

The initial PK model of choice will be a compartmental model with linear and nonlinear drug elimination. Further model testing will include, but it is not limited to, a compartmental model with target mediated drug disposition (TMDD) and a minimal PBPK model with TMDD incorporated. We anticipate TMDD to be driven by soluble LAG3 (sLAG3). However, if data allow, we plan to test also more complex models with TMDD driven by both, sLAG3 and T-cell bound LAG3.

The final PK model, possibly incorporating TMDD, will be used to develop a PK-RO model. Data relative to CD4+CD45RA- cell count will be used to model RO (quantified by J11L1 marker) and T-cell depletion (quantified by 1B4 marker). The initial RO model will likely be an Emax model. More complex models might be investigated if the data support it.

If plots (and summary) of NCA derived PK parameters identified ADA status, and/or HV vs Pso as possible significant covariates, we will investigate the influence of these covariates in the PK and RO models. Other covariates may be explored as appropriate.

#### **CONFIDENTIAL**

200630

Model acceptability will be judged by convergence, covariance estimation and standard goodness-of-fit plots that may include, but are not limited to:

- Population and individual predictions versus observations
- Conditional weighted residuals versus population predictions and time

For the final PK and the final RO models visual predictive checks (VPCs) will be conducted to assess graphically whether simulations from the developed models are able to reproduce both the central trend and variability in the observed data from the current study as a function of time.

The VPC will be based on 1000 simulations with the model and the design structure of the observed data (i.e. dose level and time, time of PK sampling and individual values of model covariates, if any). The median and the 10th and 90th will be compared to the observed data. Stratification by dose level of GSK2831781 will be used. Other stratification, such as healthy/ psoriasis will be applied in case these covariates were tested in the model.

# 14.8. Appendix 8: Abbreviations & Trade Marks

### 14.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| %AUCex | Percentage of AUC(0-¥) obtained by extrapolation |
| μg | Microgram |
| A&R | Analysis and Reporting |
| ABC | airway, breathing, and circulation from Basic Life Support |
| aCCR4 | Anti C-C chemokine receptor type 4 |
| ADA | Anti-drug antibody |
| ADA | Anti-drug antibodies |
| ADCC | Antibody Dependent Cell Cytotoxicity |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| ALT | Alanine aminotransferase (SGPT) |
| AST | Aspartate aminotransferase (SGOT) |
| AUC | Area under the concentration-time curve |
| | Area under the concentration-time curve from time zero (pre-dose) |
| $AUC(0-\infty)$ | extrapolated to infinite time |
| | Area under the concentration-time curve from time zero (pre-dose) to |
| | last time of quantifiable concentration within a subject across all |
| AUC(0-t) | treatments |
| | Area under the concentration-time curve from zero (pre-dose) to some |
| AUC(0-x) | fixed nominal time x |
| BCG | Bacillus Calmette Guérin vaccine |
| BMI | Body mass index |
| BSA | Body surface area |
| CFB | Change from baseline |
| CI | Confidence Interval |
| CL | Systemic clearance of parent drug |
| Cmax | Maximum observed concentration |
| CMV | Cytomegalovirus |
| CPK | Creatine phosphokinase |
| CPMS | Clinical Pharmacology Modelling and Simulation |
| CPR | Cardio-Pulmonary Resuscitation |
| CPSSO | Clinical Pharmacology Sciences and Study Operations |
| CRF | Case Report Form |
| CRP | C-Reactive Protein |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTLA | Cytotoxic T-Lymphocyte Antigen |
| CTR | Clinical Trial Register |
| CVb / CVw | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| CXCR | CXC Chemokine Receptor |
| DC | Dendritic Cells |

| Abbreviation | Description |
|---|---|
| DEC | Dose Escalation Committee |
| DMPK | Drug Metabolism and Pharmacokinetics |
| DOB | Date of Birth |
| DP | Decimal Places |
| DPT | Diphtheria, pertussis, tetanus |
| DTH | Delayed type hypersensitivity |
| EBV | Epstein-Barr Virus |
| ECG | Electrocardiogram |
| ECL | Immunoelectrochemiluminescent |
| eCRF | Electronic Case Record Form |
| EDTA | Ethylenediaminetetraacetic acid |
| EMA | European Medicines Agency |
| FCS | Foetal Calf Serum |
| FDA | |
| FDAAA | Food and Drug Administration |
| | Food and Drug Administration Clinical Results Disclosure Requirements |
| FTIH | First Time In Human |
| GCP | Good Clinical Practice |
| G-CSF | Granulocyte-Colony Stimulating Factor |
| GGT | Gamma glutamyltransferase |
| GI | Gastrointestinal |
| GLP | Good Laboratory Practice |
| GSK | GlaxoSmithKline |
| h | Hour |
| HBcAb | Hepatitis B core antibody |
| HBsAg | Hepatitis B surface antigen |
| Нер В | Hepatitis B |
| Hep C | Hepatitis C |
| HIV | Human Immunodeficiency Virus |
| HRT | Hormone Replacement Therapy |
| HSV | Herpes Simplex Virus |
| IA | Interim Analysis |
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonization |
| ICU | Intensive Care Unit |
| ID | Intradermal |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IEC | Independent Ethics Committee |
| IFN-γ | Interferon-gamma |
| Ig | Immunoglobulin |
| IgM | Immunoglobulin M |
| IHC | Immunohistochemistry |
| ii TAU | Immuno-Inflammation Therapeutic Area Unity |
| IL2R | Interleukin 2 Receptor |
| ILH | Immediate local hypersensitivity |

| Abbreviation | Description |
|--------------|--------------------------------------------------------|
| IMMS | International Modules Management System |
| INR | International Normalised Ratio |
| IP | Investigational Product |
| kg | Kilogram |
| L | Litres |
| LAG-3 | Lymphocyte Activation Gene 3 |
| LAG-3 | Lower Limit of Quantification |
| | ` |
| mg<br>ml | Milligram Millilitre |
| MlU/mL | milli-international units per millilitre |
| mm | Millimetre |
| MMR | Measles, mumps, rubella |
| MMRM | Mixed Model Repeated Measures |
| mRNA | Messenger Ribonucleic Acid |
| MRT | Mean Residence Time |
| NK | Natural Killer |
| nM | Nanomolar |
| NOAEL | No Observed Adverse Effect Level |
| PASI | Psoriasis Area Severity Index |
| PBMC | Peripheral Blood Mononuclear Cell |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PGA | Physicians Global Assessment |
| PK | Pharmacokinetic |
| PLSS | Plaque Lesional Severity Score |
| PPD | Tuberculin Purified Protein Derivative |
| QTc | Electrocardiogram QT interval corrected for heart rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting and Analysis Plan |
| RBC | Red blood cells |
| RNA | Ribonucleic acid |
| RO | Receptor Occupancy |
| RT-PCR | Reverse transcription polymerase chain reaction |
| SAC | Statistical Analysis Complete |
| SAE | Serious adverse event(s) |
| SGOT | Serum glutamic-oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| sLAG-3 | Soluble Lymphocyte Activation Gene 3 |
| SOP | Standard Operation Procedure |
| SPC | Summary of Product Characteristics |
| SPM | Study Procedures Manual |
| $t^{1/2}$ | Terminal phase half-life |
| TA | Therapeutic Area |
| 171 | Therapeutic Area |

| Abbreviation | Description |
|--------------|-----------------------------------------|
| TB | Tuberculosis |
| TFL | Tables, Figures & Listings |
| tlast | Time of last quantifiable concentration |
| tmax | Time of occurrence of Cmax |
| UK | United Kingdom |
| USA | United States of America |
| Vss | Volume of distribution at steady state |
| VZV | Varicella Zoster Virus |
| WBC | White blood cells |
| λz | Terminal elimination rate |

### 14.8.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| ADVAIR |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

### 14.9. Appendix 9: List of Data Displays

### 14.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|----------------|----------------|
| Study Population | 1.1 to 1.14 | Not applicable |
| Efficacy | 2.1 to 2.23 | 2.1 to 2.n |
| Safety | 3.1 to 3.35 | 3.1 to 3.6 |
| Pharmacokinetic | 4.1 to 4.6 | 4.1 to 4.6 |
| Population Pharmacokinetic (PopPK) | Not applicable | Not applicable |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.14 | 6.1 to 6.18 |
| Pharmacokinetic / Pharmacodynamic | Not applicable | Not applicable |
| Section | List | ings |
| ICH Listings | 1 to | 31 |
| Other Listings | 32 t | o 63 |

### 14.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Example Mock Shells for Data Displays.

Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' column as 'Reference.'

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

### 14.9.3. Deliverables

Following review of the IA2 and IA W2 outputs and finalisation of the database, the final list of outputs to be re-run at SAC will be reviewed.

| Delivery | Description |
|---|---|
| IA1 | Interim Analysis 1 Statistical Analysis Complete |
| IA2 EFF Interim Analysis 2 Statistical Analysis Complete for Efficacy endpoints | |
| IA2 Interim Analysis 2 Statistical Analysis Complete | |
| IA2 W2 Interim Analysis 2 Wave 2 Statistical Analysis Complete | |
| SAC | Final Statistical Analysis Complete |

# 14.9.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | • | • |
| 1.1. | safety | ES1 | Summary of subject disposition for healthy volunteers | by treatment group - 8 groups | IA1<br>IA2 W2 |
| 1.2. | safety | ES1 | Summary of subject disposition for psoriasis patients | Same as for HV - 4 groups | IA2W2 |
| 1.3. | All screened | ES6 | Summary of reasons for screen failures for healthy volunteers | Not by treatment group | SAC |
| 1.4. | All screened | ES6 | Summary of reasons for screen failures for psoriasis patients | Same as for HV | SAC |
| Protoc | ol Deviation | | | | |
| 1.5. | Safety | DV1A | Summary of important protocol deviations for healthy volunteers | by treatment group - 8 groups | SAC |
| 1.6. | Safety | DV1A | Summary of important protocol deviations for psoriasis patients | Same as for HV - 4 groups | SAC |
| Popula | ation Analysed | | | • | |
| 1.7. | All screened | SA1 | Summary of study populations for healthy volunteers | by treatment group - 8 groups See text for screen failures | IA2 W2 |
| 1.8. | All<br>screened | SA1 | Summary of study populations for psoriasis patients | Same as for HV - 4 groups<br>See text for screen failures | IA2 W2 |

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Demog | raphic and Bas | eline Characteris | tics | | • |
| 1.9. | safety | DM1 | Summary of demographic characteristics for healthy volunteers | <ol> <li>by treatment group - 8 groups</li> <li>Include: Gender, height, weight and BMI</li> <li>Include age category: &lt;18 years, 18 to 65 years, 66 to 75 years and &gt;75 years</li> </ol> | IA2 W2 |
| 1.10. | safety | DM1 | Summary of demographic characteristics for psoriasis patients | Same as for HV - 4 groups | IA2 W2 |
| 1.11. | safety | DM5 | Summary of race and racial combinations for healthy volunteers | <ol> <li>by treatment group - 8 groups</li> <li>Report only categories where n&gt;0 count</li> </ol> | SAC |
| 1.12. | safety | DM5 | Summary of race and racial combinations for psoriasis patients | Same as for HV - 4 groups | SAC |
| 1.13. | safety | DM11 | Summary of age ranges for healthy volunteers | by treatment group - 8 groups | SAC |
| 1.14. | safety | DM11 | Summary of age ranges for psoriasis patients | by treatment group - 4 groups | SAC |

# 14.9.5. Efficacy Tables

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DTH inc | duration | | | | |
| 2.1. | Safety | | Summary of induration diameter for healthy volunteers (DTH subjects) | <ol> <li>Absolute and CFB</li> <li>by challenge site (4) and overall =&gt; 5 parameters</li> <li>2 treatment groups (cohort</li> <li>placebo (DTH) and 0.15mg (DTH=ADA-ve)</li> </ol> | IA1 |
| 2.2. | Safety | | Summary results of statistical analysis of change from baseline in induration diameter for healthy volunteers (DTH subjects) | 1. for overall only (1 parameter) 3. 2 treatment groups (cohort 5): placebo (DTH) and 0.15mg (DTH=ADA-ve) | IA1 |
| 2.3. | safety | | Summary of duration of induration for healthy volunteers (DTH subjects) | 1. Absolute 2. 2 treatment groups: placebo (DTH) and 0.15mg (DTH=ADA-ve) 3. If needed for SAC, include only the summary of observed duration (no HR estimate) | IA1 |
| BSA | | | | | |
| 2.4. | Safety | | Summary of body surface area by visit for psoriasis patients | <ol> <li>Absolute, CFB, %CFB</li> <li>4 regional BSA</li> <li>Total BSA (sum of the 4 regional BS)</li> </ol> | SAC |

| Efficac | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PASI | | | | | |
| 2.5. | Safety | TE1 | Summary of PASI scores by visit for psoriasis patients | <ol> <li>By treatment group - 4<br/>groups</li> <li>Absolute, CFB, %CBF (byline)</li> </ol> | IA2 EFF |
| 2.6. | Safety | TE2 | Summary of PASI50 and PASI75 responders by visit for psoriasis patients | <ol> <li>By treatment group - 4 groups</li> <li>PASI50/75</li> <li>Footnote: PASI50 or PASI75 responders are patients with a ≥ 50% or 75% reduction in PASI score from baseline</li> </ol> | IA2 EFF |
| 2.7. | Safety | TE3 | Summary of statistical analysis results for change from baseline in PASI scores over time for psoriasis patients | | IA2 EFF |
| PLSS | | | | | |
| 2.8. | Safety | TE1 | Summary of PLSS scores by visit for psoriasis patients | <ol> <li>Same table as for PASI</li> <li>Index and biospy lesions<br/>(byline)</li> <li>Absolute, CFB, %CBF (byline)</li> </ol> | IA2 EFF |
| 2.9. | Safety | TE3 | Summary of statistical analysis results for change from baseline in PLSS scores over time for psoriasis patients | <ol> <li>Same as for PASI</li> <li>Index lesion only</li> <li>CFB</li> </ol> | IA2 EFF |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PGA | | | | | |
| 2.10. | Safety | TE1 | Summary of PGA scores by visit for psoriasis patients | <ol> <li>Absolute, CFB</li> <li>Considers categories as continuous</li> </ol> | IA2 EFF |
| 2.11. | Safety | TE2 | Summary of PGA responders by visit for psoriasis patients | Same table as for PASI50/75 (include exact CI) Footnote: definition of PGA responders | IA2 EFF |
| 2.12. | Safety | TE4 | Summary of PGA responses by visit for psoriasis patients | Frequency count (categorical variable) | IA2 EFF |
| Endpoi | nts for go/no g | o decisions | | | |
| 2.13. | Safety | | Bayesian analyses of key endpoints | See Section 13 IA2 EFF: PASI and PLSS IA2: total LAG3 cells, Ki67, epidermis thickness Need to add SAS log + CV plots | IA2 EFF<br>IA2 |

# 14.9.6. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DTH in | duration | | | | |
| | | | | <ol> <li>Absolute</li> <li>by challenge site (4) and overall =&gt; 5 parameters</li> </ol> | |
| 2.1. | safety | safety F_PD1 | Individual plot of induration diameter over time for healthy volunteers (DTH subjects) | 3. 2 treatment groups (cohort 5): placebo (DTH) and 0.15mg (DTH=ADA-ve) | IA1 |
| | | | | 4. ADA+ve subjects identified in legend | |
| 2.2. | safety | safety F_PD3 | Mean ( $\pm$ SD) induration diameter over time for healthy volunteers (DTH subjects) | <ol> <li>Absolute</li> <li>by challenge site (4) and overall =&gt; 5 parameters -</li> <li>2 treatment groups (cohort</li> </ol> | IA1 |
| | | | | 5): placebo (DTH) and 0.15mg<br>(DTH=ADA-ve) | |
| | safety | | Adjusted mean (95% CI) of change from baseline in | 1. CFB (LS means) 2. overall only | |
| 2.3. | | safety | safety F_ | ety F_PD3 induration diameter over time for healthy volunteers (DTH subjects) | 3. 2 treatment groups (cohort 5): placebo (DTH) and 0.15mg (DTH=ADA-ve) |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PASI | | | | | |
| 2.4. | Safety | F_PD1 | Individual plot of PASI scores over time for psoriasis patients | <ol> <li>Absolute and %CFB</li> <li>ADA+ve subjects identified in legend</li> </ol> | IA2 EFF |
| 2.5. | Safety | F_PD3 | Mean (±SD) PASI scores over time for psoriasis patients | Absolute, %CFB | IA2 EFF |
| 2.6. | Safety | F_PD3 | Adjusted mean (95% CI) of change from baseline in PASI scores over time for psoriasis patients | CFB | IA2 EFF |
| PLSS | • | | | | |
| 2.7. | Safety | F_PD1 | Individual plot of PLSS scores over time for psoriasis patients | <ol> <li>Absolute and %CFB</li> <li>Index and biospy lesions</li> <li>ADA+ve subjects identified in legend</li> </ol> | IA2 EFF |
| 2.8. | Safety | F_PD3 | Mean (±SD) PLSS scores over time for psoriasis patients | Absolute, %CFB Index lesion only | IA2 EFF |
| 2.9. | Safety | F_PD3 | Adjusted mean (95% CI) of change from baseline in PLSS scores over time for psoriasis patients | CFB<br>Index lesion only | IA2 EFF |
| PGA | | | | | |
| 2.10. | Safety | F_PD1 | Individual plot of PGA responses over time for psoriasis patients | <ol> <li>Absolute only</li> <li>Considers categories as continuous</li> <li>ADA+ve subjects identified in legend</li> </ol> | IA2 EFF |

# 14.9.7. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AEs) | | | | |
| 3.1. | safety | CP_AE1P | Summary of all adverse events for healthy volunteers | <ol> <li>by treatment group - 9 groups (including total active)</li> <li>Only TEAE</li> <li>by SOC then PT</li> <li>Notes:</li> <li>Total Active: Total over the 5 doses (except Placebo for HV Combined).</li> <li>ADA status as defined at screening.</li> <li>Combined treatment groups include subjects with ADA-ve and ADA+ve.</li> <li>Only treatment-emergent AEs are summarised: starting date between 1st dose and last scheduled visit (follow-up or combined FU/surveillance)</li> </ol> | IA1<br>IA2 W2 |
| 3.2. | safety | CP_AE1P | Summary of all adverse events for psoriasis patients | Same as for HV - 5 groups (including total active) | IA2 W2 |
| 3.3. | safety | CP_AE1P | Summary of drug-related adverse events for healthy volunteers | same output as for all AEs | IA1<br>IA2 W2 |
| 3.4. | safety | CP_AE1P | Summary of drug-related adverse events for psoriasis patients | Same as for HV - 5 groups (including total active) | IA2 W2 |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.5. | safety | CP_AE1P | Summary of all adverse events for ADA+ve subjects | 1. ADA+ve defined as subject who were ADA+ve at screening visit 2. Parts A and B (cohorts 5, 7-9) => groups: Pbo HV, 0.15mg/kg, Pbo PsO, 0.5mg/kg, 1.5mg/kg, 5mg/kg 3. Only TEAE 4. by SOC then PT | SAC |
| 3.6. | safety | AE3 | Summary of common adverse events for healthy volunteers | 1. Common defined as at least 2 patients with the event in any of the treatment groups, separately for parts A and B 2. by treatment group - 9 groups (including total active) 3. Only TEAE 4. by PT | IA2 W2 |
| 3.7. | safety | AE3 | Summary of common adverse events for psoriasis patients | Same as for HV - 5 groups (including total active) | IA2 W2 |
| 3.8. | safety | CP_AE1P | Summary of all adverse events (healthy volunteers and psoriasis patients) | Same as for HV or PsO Include 4 columns - Placebo for HV - Total Active (HV) - Placebo for PsO - Total active (PsO) | IA2 W2 |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.9. | safety | AE2 | Relationship between system organ class and verbatim text | HV and PsO in the same summary table | SAC |
| Serious | Serious Adverse Events | | | | |
| 3.10. | safety | AE1 | Summary of serious adverse events for healthy volunteers | <ol> <li>by treatment group - 9<br/>groups (including total active)</li> <li>Only TEAE</li> <li>by PT</li> </ol> | IA1<br>IA2 W2 |
| 3.11. | safety | AE1 | Summary of serious adverse events for psoriasis patients | Same as for HV - 5 groups (including total active) | IA2 W2 |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Labora | tory: Chemistry | y | | | |
| 3.12. | safety | LB1 | Summary of chemistry by visit for healthy volunteers | <ol> <li>by treatment group - 8 groups</li> <li>By visit, from baseline to last scheduled visit (excluding surveillance visit)</li> </ol> | IA1<br>IA2 W2 |
| 3.13. | safety | LB1 | Summary of chemistry by visit for psoriasis patients | Same as for HV - 4 groups | IA2 W2 |
| 3.14. | safety | LB3 | Summary of change from baseline in chemistry by visit for healthy volunteers | <ol> <li>by treatment group - 8<br/>groups</li> <li>All post-baseline visits,<br/>excluding surveillance visits</li> </ol> | IA1<br>SAC |
| 3.15. | safety | LB3 | Summary of change from baseline in chemistry by visit for psoriasis patients | Same as for HV - 4 groups | SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.16. | safety | LB1 | Summary of haematology by visit for healthy volunteers | same output as for chemistry parameters | IA1<br>IA2 W2 |
| 3.17. | safety | LB1 | Summary of haematology by visit for psoriasis patients | same output as for chemistry parameters | IA2 W2 |
| 3.18. | safety | LB3 | Summary of change from baseline in haematology by visit for healthy volunteers | same output as for chemistry parameters | IA1<br>SAC |
| 3.19. | safety | LB3 | Summary of change from baseline in haematology by visit for psoriasis patients | same output as for chemistry parameters | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Laborat | tory: Urinalysis | <b>.</b> | | | |
| 3.20. | safety | UR3 | Summary of urinalysis dipstick results by visit for healthy volunteers | <ol> <li>by treatment group - 8<br/>groups</li> <li>By visit, from screening to last<br/>scheduled visit (excluding<br/>surveillance visit)</li> </ol> | IA1<br>SAC |
| 3.21. | safety | UR3 | Summary of urinalysis dipstick results by visit for psoriasis patients | Same as for HV - 4 groups | SAC |
| ECG | | | | | |
| 3.22. | safety | EG1 | Summary of ECG findings by visit for healthy volunteers | 1. by treatment group - 8 groups 2. By visit, from screening to last scheduled visit (excluding surveillance visit) 3. For screening, use the worst finding out of the 3 values – add the following footonote for screening visit only: At screening, the finding for a subject is the worst finding observed across the 3 findings. | IA1<br>IA W2 |
| 3.23. | safety | EG1 | Summary of ECG findings by visit for psoriasis patients | Same as for HV - 4 groups | IA W2 |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.24. | safety | EG2 | Summary of ECG values by visit for healthy volunteers | <ol> <li>by treatment group - 8 groups</li> <li>By visit, from baseline to last scheduled visit (excluding surveillance visit)</li> </ol> | SAC |
| 3.25. | safety | EG2 | Summary of ECG values by visit for psoriasis patients | Same as for HV - 4 groups | SAC |
| 3.26. | safety | EG2 | Summary of change from baseline in ECG values by visit for healthy volunteers | by treatment group - 8 groups | SAC |
| 3.27. | safety | EG2 | Summary of change from baseline in ECG values by visit for psoriasis patients | Same as for HV - 4 groups | SAC |
| 3.28. | safety | EG10/EG11<br>combined | Summary of maximum emergent QTc values by category (absolute and change from baseline) for healthy volunteers | Includes baseline values, and footnote: note: the maximum change for a subject is the maximum increase from baseline observed across all time points for the subject | SAC |
| 3.29. | safety | EG10/EG11 combined | Summary of maximum emergent QTc values by category (absolute and change from baseline) for psoriasis patients | Same as for HV - 4 groups | SAC |
| Vital Si | gns | | | | |
| 3.30. | safety | VS1 | Summary of vital signs by visit for healthy volunteers | <ol> <li>by treatment group - 8<br/>groups</li> <li>Include the temperature</li> </ol> | IA1<br>IA2 W2 |
| 3.31. | safety | VS1 | Summary of vital signs by visit for psoriasis patients | Same as for HV - 4 groups | IA2 W2 |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.32. | safety | VS1 | Summary of change from baseline in vital signs by visit for healthy volunteers | Same as for absolute values | SAC |
| 3.33. | safety | VS1 | Summary of change from baseline in vital signs by visit for psoriasis patients | Same as for HV - 4 groups | SAC |
| Cytokir | ies | | | | |
| 2.24 | Safety | Safety | Summary of cytokines for healthy volunteers | 1. Absolute, CFB | IA1 |
| 3.34. | | | | 2. See parameters in RAP text | SAC |
| 3.35. | Safety | | Summary of cytokines for psoriasis patients | Same as HV | IA2 |
| Advers | e events (addit | ional) | | | |
| 3.36. | Safety | CP_AE1P | Summary of drug-related adverse events for healthy volunteers and psoriasis patients | Same as for HV or PsO only For HV, remove combined 0.15mg/kg (only keep separate ADA status | SAC |
| 3.37. | Safety | CP_AE1P | Summary of all adverse events for healthy volunteers and psoriasis patients | Same as for HV or PsO only For HV, remove combined 0.15mg/kg (only keep separate ADA status | SAC |

| Safety: | afety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Immun | ophenotyping | | | | |
| 3.38. | Safety | | Summary of immunophenotyping for healthy volunteers | Same output as for flow cytometry for the following parameters. For the 4 of them concentration should be used. No derivation is needed. marker code / marker / endpoint: CDX219 / CD45+ CD3+ / Pan T cells CDX220 / CD45+ CD3+ CD8+ / CD8 T cells CDX221 / CD45+ CD3+ CD8- / CD4 T cells CDX225 / CD45+ CD3- CD16+ CD56+ / NK cells | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.39. | Safety | | Summary of immunophenotyping for psoriasis patients | Same output as for flow cytometry for the following parameters. For the 4 of them concentration should be used. No derivation is needed. marker code / marker / endpoint: CDX219 / CD45+ CD3+ / Pan T cells CDX220 / CD45+ CD3+ CD8+ / CD8 T cells CDX221 / CD45+ CD3+ CD8- / CD4 T cells CDX225 / CD45+ CD3- CD16+ CD56+ / NK cells | SAC |

# 14.9.8. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Labora | tory | | | | |
| 3.1. | safety | LB11 | Individual plot of lymphocytes and neutrophils over time for healthy volunteers | <ol> <li>panel per treatment group - 8 groups</li> <li>ADA+ve subjects identified in legend</li> </ol> | SAC |
| 3.2. | safety | LB11 | Individual plot of lymphocytes and neutrophils over time for psoriasis patients | Same as for HV - 4 groups | SAC |
| ECG | • | | | | |
| 3.3. | safety | EG7 | Empirical distribution function for maximum increase from baseline in QTcF interval for healthy volunteers | <ol> <li>8 treatment groups on one plot</li> <li>Calculate the maximum change from baseline</li> </ol> | SAC |
| 3.4. | safety | EG7 | Empirical distribution function for maximum increase from baseline in QTcF interval for psoriasis patients | Same as for HV - 4 groups | SAC |
| 3.5. | safety | EG7 | Empirical distribution function for maximum increase from baseline in QTcB interval for healthy volunteers | Same as QTcF | SAC |
| 3.6. | safety | EG7 | Empirical distribution function for maximum increase from baseline in QTcB interval for psoriasis patients | Same as for HV - 4 groups | SAC |
| lmmur | nophenotyping | g | | | |
| 3.7. | Safety | | Individual plot of immunophenotyping over time for healthy volunteers | Same plot as for key flow parameters (see Figure 6.8) | SAC |
| 3.8. | Safety | | Individual plot of immunophenotyping over time for psoarisis patients | Same plot as for key flow parameters (see Figure 6.9) | SAC |
#### 14.9.9. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PK cor | centration | | | | |
| 4.1. | PK | PK01 | Summary of plasma GSK2831781 pharmacokinetic concentration-time data for healthy volunteers | by treatment group - 7 groups (placebo not included) Remove 95%CI as not normally distributed | IA2 W2 |
| 4.2. | PK | PK01 | Summary of plasma GSK2831781 pharmacokinetic concentration-time data for psoriasis patients | same as HV – 3 groups (placeo not included) | IA2 W2 |
| PK der | ived parameter | S | | | |
| 4.3. | PK | PK03 | Summary of derived plasma GSK2831781 pharmacokinetic parameters for healthy volunteers | by treatment group - 7 groups (placebo not included) | IA2 W2 |
| 4.4. | PK | PK03 | Summary of derived plasma GSK2831781 pharmacokinetic parameters for psoriasis patients | same as HV – 3 groups (placeo not included) | IA2 W2 |
| 4.5. | PK | PK05 | Summary of log-transformed derived plasma<br>GSK2831781 pharmacokinetic parameters for healthy<br>volunteers | by treatment group - 7 groups (placebo not included)¶ Exclude tmax and tlast | IA2 W2 |
| 4.6. | PK | PK05 | Summary of log-transformed derived plasma<br>GSK2831781 pharmacokinetic parameters for psoriasis<br>patients | same as HV – 3 groups (placeo not included) | IA2 W2 |

# 14.9.10. Pharmacokinetic Figures

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| PK con | centration | | | | |
| 4.1. | PK | PK24 | Individual GSK2831781 plasma concentration-time plot (linear and semi-log) for healthy volunteers | <ol> <li>by treatment group - 8 groups</li> <li>Treatment group as page variable</li> <li>x-axis displays actual relative time.</li> <li>Include line for LLQ along with footnote defining LLQ value</li> <li>ADA +ve patients identified in legend</li> </ol> | IA2 W2 |
| 4.2. | PK | PK24 | Individual GSK2831781 plasma concentration-time plot (linear and semi-log) for psoriasis patients | Same as for HV - 4 groups | IA2 W2 |
| 4.3. | PK | PK17 | Mean plasma GSK2831781 concentration-time plots (linear and semi-log) for healthy volunteers | <ol> <li>by treatment group - 7 groups (placebo not included)3. x-axis displays actual relative time.</li> <li>Same y-axis for HV and PsO</li> <li>Include line for LLQ along with footnote defining LLQ value</li> </ol> | IA2 W2 |
| 4.4. | PK | PK17 | Mean plasma GSK2831781 concentration-time plots (linear and semi-log) for psoriasis patients | same as for HV | IA2 W2 |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PK deri | ved parameter | S | | , | |
| 4.5. | PK | PK28 | Individual GSK2831781 pharmacokinetic parameters versus dose for healthy volunteers | 1. For Cmax, AUC[0-last] - Parameters as page variable 2. x-axis: 5 doses (0.15 combined) 4. ADA +ve patients identified in legend | IA2 W2 |
| 4.6. | PK | PK28 | Individual GSK2831781 pharmacokinetic parameters versus dose for psoriasis patients | Same as for HV - 3 doses | IA2 W2 |

# 14.9.11. Pharmacodynamic / Biomarker Tables

| | | . DSL / DSL / | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable |
| IHC pa | rameters | • | | | |
| 6.1. | Safety | | Summary of LAG3+ and CD3+ in skin by visit for healthy volunteers (DTH subjects) | 1. Absolute, CFB, %CFB 2. 2 visits: baseline and day 4 3. Endpoints: CD3+, LAG3+ (check RAP text) 4. 2 treatment groups: placebo (DTH) and 0.15mg (DTH=ADA-ve) | IA1<br>IA2 |
| 6.2. | Safety | | Summary of cells in lesional biopsies measured by IHC by visit for psoriasis patients | <ol> <li>Results for dermis and epidermis for CD3+, lag3+; epidermis only for Ki67</li> <li>Absolute, CFB, %CFB</li> <li>2 visits: baseline and day 29</li> <li>4 treatment groups</li> </ol> | IA2 |
| 6.3. | Safety | | Summary of epidermis thickness by visit for psoriasis patients | Same as for IHC parameters | IA2 |
| 6.4. | Safety | | Summary of statistical analysis results for change from baseline in LAG3+ and CD3+ values for healthy volunteers (DTH subjects) | 1. CFB 2. Endpoints: CD3+, LAG3+ (check RAP text) 3. 2 treatment groups: placebo (DTH) and 0.15mg (DTH=ADA-ve) | IA1<br>IA2 |

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.5. | Safey | | Summary of statistical analysis results for change from baseline in cells in lesional biopsies measured by IHC for psoriasis patients | 1. Results for dermis and epidermis for CD3+, lag3+; epidermis only for Ki67 and epidermis thickness 2. CFB 3. 4 treatment groups | IA2 |
| Flow cy | tometry | | | <u> </u> | |
| 6.6. | Safety | | Summary of flow cytometry by visit for healthy volunteers | 1. Only the 6 key flow parameters - see RAP text 2. Absolute, CFB, % of baseline | IA1<br>IA2 |
| 6.7. | Safety | | Summary of flow cytometry by visit for psoriasis patients | Same as for HV | IA2 |
| s-LAG3 | | | | | |
| 6.8. | Safety | | Summary of sLAG-3 by visit for healthy volunteers | 1. Absolute, CFB | IA1<br>IA2 |
| 6.9. | Safety | | Summary of sLAG-3 by visit for psoriasis patients | Same as for HV | IA2 |
| Immun | ogenicity | <u>'</u> | | | |
| 6.10. | Safety | IMM1 | Summary of positive immunogenicity results for healthy volunteers | | IA1<br>IA2 W2 |
| 6.11. | Safety | IMM1 | Summary of positive immunogenicity results for psoriasis patients | Same as for HV | IA2 W2 |

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Transc | riptomics | | | | • |
| 6.12. | Safety | | Summary of blood transcriptomics for healthy volunteers | (same mockshell as for any efficacy endpoint, e.g. pasi) By gene (2 as not housekeeping genes) and summary (delta delta Ct and fold change) | SAC |
| 6.13. | Safety | | Summary of blood transcriptomics for psoriasis patients | Same as for HV | SAC |
| 6.14. | Safety | | Summary of biopsy transcriptomics for psoriasis patients | Same as for blood<br>transcriptomics<br>No data for HV<br>Displays visit 15 (only cohort 7 –<br>3 on placebo, 6 on 0.5mg/kg)<br>and Day 29 (all PSO) | IA2 W2 (as issue with mapping program from raw data to SI data – 3 gene codes missing) |

# 14.9.12. Pharmacodynamic / Biomarker Figures

| Pharma | Pharmacodynamic and Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| IHC par | ameters | | | | |
| 6.1. | Safety | F_PD1 | Individual plot of LAG3+ and CD3+ in skin over time for healthy volunteers (DTH subjects) | <ol> <li>Absolute and CFB</li> <li>Total cells (HPF 1-5) - average across 3 skin layers (check RAP text)</li> <li>2 visits: baseline and day 4</li> <li>Endpoints: CD3+, lag3+</li> </ol> | IA1<br>IA2 |
| 6.2. | Safety | F_PD1 | Individual plot of cells in lesional biopsies measured by IHC over time for psoriasis patients | <ol> <li>Results for dermis and epidermis for CD3+ and lag3+; epidermis only for Ki67</li> <li>Absolute and CFB</li> <li>2 visits: baseline and day 29</li> <li>Endpoints: CD3+, lag3+, Ki67, (seprate table as different dataset)</li> <li>See RAP text for endpoints</li> </ol> | IA2 |
| 6.3. | Safety | F_PD1 | Individual plot of epidermis thickness over time for psoriasis patients | Same as for IHC endpoints | IA2 |

| Pharma | Pharmacodynamic and Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.4. | Safety | F_PD2 | Subject profiles of LAG3+ and CD3+ in skin for healthy volunteers (DTH subjects) | 1. LAG3+, CD3+ (check RAP text) 2. 2 treatment groups: placebo (DTH) and 0.15mg (DTH=ADA-ve) 3. Total number of cells per layer (3) + average => 4 lines per subjects 4. Absolute 5. Panel with subjects 6. Footnote to be added | IA1<br>IA2 |
| 6.5. | Safety | F_PD3 | Mean (±SD) LAG3+ and CD3+ in skin over time for healthy volunteers(DTH subjects) | 1. LAG3+, CD3+ (check RAP text) Only average 2. 2 treatment groups: placebo (DTH) and 0.15mg (DTH=ADA-ve) 3. Absolute | IA1<br>IA2 W2 |
| 6.6. | Safety | F_PD3 | Mean (±SD) cells in lesional biopsies measured by IHC over time for psoriasis patients | <ol> <li>Results for dermis and epidermis for CD3+, lag3+; epidermis only for Ki67</li> <li>Absolute</li> <li>2 visits: baseline and day 29</li> <li>Endpoints: CD3+, lag3+, Ki67</li> <li>4 treatment groups</li> </ol> | IA2 W2 |
| 6.7. | Safety | F_PD3 | Mean (±SD) epidermis thickness over time for psoriasis patients | Same as for IHC endpoints | IA2 W2 |

| Pharma | Pharmacodynamic and Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Flow cy | tometry | | | | |
| 6.8. | Safety | F_PD1 | Individual plot of flow cytometry key parameters over time for healthy volunteers | <ol> <li>Only the 6 key flow parameters - see RAP text</li> <li>Absolute, % of baseline</li> <li>ADA+ve subjects identified in legend</li> </ol> | IA1<br>IA2 |
| 6.9. | Safety | F_PD1 | Individual plot of flow cytometry key parameters over time for psoriasis patients | Same as for HV | IA2 |
| 6.10. | Safety | F_PD3 | Mean (±SD) flow cytometry key parameters over time for healthy volunteers | 1. Only the 6 key flow parameters - see RAP 2. % of baseline | IA2 |
| 6.11. | Safety | F_PD3 | Mean (±SD) flow cytometry key parameters over time for psoriasis patients | Same as for HV | IA2 |
| s-LAG3 | } | | | | |
| 6.12. | Safety | F_PD1 | Individual plot of s-LAG3 over time for healthy volunteers | Absolute, CFB ADA+ve subjects identified in legend | IA1<br>IA2 |
| 6.13. | Safety | F_PD1 | Individual plot of s-LAG3 over time for psoriasis patients | Same as for HV | IA2 |
| 6.14. | Safety | F_PD3 | Mean (±SD) s-LAG3 over time for healthy volunteers | CFB | IA2 W2 |
| 6.15. | Safety | F_PD3 | Mean (±SD) s-LAG3 over time for psoriasis patients | Same as for HV | IA2 W2 |

| Pharma | Pharmacodynamic and Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Transc | riptomics | | | | |
| 6.16. | Safety | F_PD4 | Boxplot of the blood transcriptomics for healthy volunteers | 1. By gene (not including housekeeping genes) and summary (delta delta Ct and fold change) - only 1 visit Day 2 2. x-axis: treatment group 3. Individual values (jittered) displayed on top of the boxplot 4. Add footnote about the values in the boxplot | SAC |
| 6.17. | Safety | F_PD4 | Boxplot of the blood transcriptomics for psoriasis patients | Same as for HV | SAC |
| 6.18. | Safety | F_PD4 | Boxplot of the biopsy transcriptomics for psoriasis patients | Same as for HV Display only versus Day 29 (not day 15) | IA2 W2 |
| Flow cy | tometry | | | | |
| 6.19. | Safety | F_PD3 | Mean (±SE) flow cytometry key parameters up to Day 29 Visit for healthy volunteers | 1. Only the 6 key flow parameters - see RAP 2. % of baseline | SAC |
| 6.20. | Safety | F_PD3 | Mean (±SE) flow cytometry key parameters up to Day 29<br>Visit for psoriasis patients | 1. Only the 6 key flow parameters - see RAP 2. % of baseline | SAC |
| s-LAG3 | | | | | |
| 6.21. | Safety | F_PD3 | Mean (±SD) s-LAG3 up to Day 29 Visit for healthy volunteers | СҒВ | SAC |

| Pharmacodynamic and Biomarker: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.22. | Safety | F_PD3 | Mean (±SD) s-LAG3 up to Day 29 Visit for psoriasis patients | CFB | SAC |

# **14.9.13.** ICH Listings

| ICH: Lis | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1. | Safety | DM2 | Listing of demographic characteristics for healthy volunteers | | IA1 |
| 2. | Safety | DM2 | Listing of demographic characteristics for psoriasis patients | | IA2 W2 |
| 3. | Safety | AE7 | Listings of subject numbers for individual adverse events for healthy volunteers | | SAC |
| 4. | Safety | AE7 | Listings of subject numbers for individual adverse events for psoriasis patients | same as for HV | IA2 W2 |
| 5. | Safety | CP_AE8 | Listing of all adverse events for healthy volunteers | | IA2 W2 |
| 6. | Safety | CP_AE8 | Listing of all adverse events for psoriasis patients | same as for HV | IA2 W2 |
| 7. | Safety | CP_AE8a | Listing of serious adverse events for healthy volunteers | Same as for all Aes | IA2 W2 |
| 8. | Safety | CP_AE8a | Listing of serious adverse events for psoriasis patients | same as for HV | IA2 W2 |
| 9. | Safety | CP_AE8 | Listing of adverse events leading to withdrawal from study for healthy volunteers | | SAC |
| 10. | Safety | CP_AE8 | Listing of adverse events leading to withdrawal from study for psoriasis patients | | SAC |
| 11. | Safety | CP_LB5 | Listing of clinical chemistry abnormalities of potential clinical importance for healthy volunteers | | IA2 W2 |
| 12. | Safety | CP_LB5 | Listing of clinical chemistry abnormalities of potential clinical importance for psoriasis patients | | IA2 W2 |
| 13. | Safety | CP_LB6 | Listing of all clinical chemistry laboratory data for subjects with PCI abnormalities for healthy volunteers | | IA1<br>SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 14. | Safety | CP_LB6 | Listing of all clinical chemistry laboratory data for subjects with PCI abnormalities for psoriasis patients | | IA2 W2 |
| 15. | Safety | CP_LB5 | Listing of haematology abnormalities of potential clinical importance for healthy volunteers | | IA2 W2 |
| 16. | Safety | CP_LB5 | Listing of haematology abnormalities of potential clinical importance for psoriasis patients | | IA2 W2 |
| 17. | Safety | CP_LB6 | Listing of all haematology laboratory data for subjects with PCI abnormalities for healthy volunteers | | SAC |
| 18. | Safety | CP_LB6 | Listing of all haematology laboratory data for subjects with PCI abnormalities for psoriasis patients | | IA2 W2 |
| 19. | Safety | UR2a | Listing of urinalysis data for healthy volunteers | | IA1<br>SAC |
| 20. | Safety | UR2a | Listing of urinalysis data for psoriasis patients | | SAC |
| 21. | Safety | | Listing of CMV and EBV serology for healthy volunteers | | SAC |
| 22. | Safety | | Listing of CMV and EBV serology for psoriasis patients | | SAC |
| 23. | Safety | CP_EG3 | Listing of ECG values of potential clinical importance for healthy volunteers | | IA2 W2 |
| 24. | Safety | CP_EG3 | Listing of ECG values of potential clinical importance for psoriasis patients | | IA2 W2 |
| 25. | Safety | CP_EG3 | Listing of all ECG values for subjects with any value of potential clinical importance for healthy volunteers | | IA2 W2 |
| 26. | Safety | CP_EG3 | Listing of all ECG values for subjects with any value of potential clinical importance for psoriasis patients | | IA2 W2 |
| 27. | Safety | CP_EG5 | Listing of abnormal ECG findings for psoriasis patients | | IA2 W2 |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 28. | Safety | CP_VS4 | Listing of vital signs of potential clinical importance for healthy volunteers | | IA2 W2 |
| 29. | Safety | CP_VS4 | Listing of vital signs of potential clinical importance for psoriasis patients | | IA2 W2 |
| 30. | Safety | CP_VS4 | Listing of all vital signs for subjects with any value of potential clinical importance for healthy volunteers | | IA1<br>SAC |
| 31. | Safety | CP_VS4 | Listing of all vital signs for subjects with any value of potential clinical importance for psoriasis patients | | SAC |
| 64 | Safety | CP_TA1 | Listing of randomised and actual treatments for healthy volunteers | | SAC |
| 65 | Safety | CP_TA1 | Listing of randomised and actual treatments for psoriasis patients | | SAC |
| 66 | Safety | ES2 | Listing of reasons for study withdrawal for healthy volunteers | | SAC |
| 67 | Safety | ES2 | Listing of reasons for study withdrawal for psoriasis patients | | SAC |
| 68 | All screened | ES7 | Listing of reasons for screening failure for healthy volunteers | | SAC |
| 69 | All screened | ES7 | Listing of reasons for screening failure for psoriasis patients | | SAC |
| 70 | Safety | DV2 | Listing of important protocol deviations for healthy volunteers | | SAC |
| 71 | Safety | DV2 | Listing of important protocol deviations for psoriasis patients | | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 72 | Safety | | Listing of Subjects with Inclusion/Exclusion Criteria Deviations for Healthy Volunteers | | SAC |
| 73 | Safety | | Listing of Subjects with Inclusion/Exclusion Criteria Deviations for Psoarisis Patients | | SAC |
| 74 | Safety | | Listing of Race for Healthy Volunteers | | SAC |
| 75 | Safety | | Listing of Race for Psoarisis Patients | | SAC |
| 76 | Safety | SA3a | Listing of subjects excluded from any population for healthy volunteers | | SAC |
| 77 | Safety | SA3a | Listing of subjects excluded from any population for psoriasis patients | | SAC |
| 78 | Safety | CP_CM3 | Listing of concomitant medications by generic term for healthy volunteers | | SAC |
| 79 | Safety | CP_CM3 | Listing of concomitant medications by generic term for psoarisis patients | | SAC |
| 80 | Safety | CP_EG5 | Listing of abnormal ECG findings for healthy volunteers | | SAC |

# 14.9.14. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 32. | PK | PK07 | Listing of plasma GSK2831781 pharmacokinetic concentration-time data for healthy volunteers | | IA2 W2 |
| 33. | PK | PK07 | Listing of plasma GSK2831781 pharmacokinetic concentration-time data for psoriasis patients | | IA2 W2 |
| 34. | PK | PK13 | Listing of derived plasma GSK2831781 pharmacokinetic parameters for healthy volunteers | | IA2 W2 |
| 35. | PK | PK13 | Listing of derived plasma GSK2831781 pharmacokinetic parameters for psoriasis patients | | IA2 W2 |
| 36. | Safety | IMM2 | Listing of immunogenicity results for healthy volunteers | NAB assay results included for SAC | IA2 W2 |
| 37. | Safety | IMM2 | Listing of immunogenicity results for psoriasis patients | same as for HV | IA2 W2 |
| 38. | Safety | | Listing of induration diameter for healthy volunteers (DTH subjects) | | IA1 |
| 39. | Safety | | Listing of duration of induration for healthy volunteers (DTH subjects) | | IA1 |
| 40. | safety | | Raw sas output statistical analysis results of change from baseline in induration diameter for healthy volunteers (DTH subjects) | | IA1 |
| 41. | safety | | Raw sas output statistical analysis results of duration of induration for healthy volunteers (DTH subjects) | | IA1 |
| 42. | Safety | LS1 | Listing of PASI-related endpoints for psoriasis patientss | | SAC |
| 43. | Safety | | Listing of PASI components for psoriasis patients | | SAC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 44. | Safety | | Listing of BSA scores for psoriasis patients | | SAC |
| 45. | Safety | | Raw sas output of statistical analysis results for change from baseline in PASI scores for psoriasis patients | | IA2 EFF<br>IA2 |
| 46. | Safety | | Raw sas output of statistical analysis results for change from baseline in PLSS score for psoriasis patients | | IA2 EFF<br>IA2 |
| 47. | Safety | | Listing of PLSS-related endpoints for psoriasis patients | | SAC |
| 48. | Safety | | Listing of PGA-related endpoints for psoriasis patients | | SAC |
| 49. | Safety | | Listing of cytokines for healthy volunteers | | IA1 |
| 50. | Safety | | Listing of cytokines for psoriasis patients | | SAC |
| 51. | Safety | | Listing of flow cytometry for healthy volunteers | All the parameters, not only the 6 key ones | IA1 |
| 52. | Safety | | Listing of flow cytometry for psoriasis patients | All the parameters, not only the 6 key ones | SAC |
| 53. | Safety | | Listing of LAG3+ and CD3+ in skin for healthy volunteers (DTH subjects) | | IA1 |
| 54. | Safety | | Listing of cells in lesional biopsies measured by IHC for psoriasis patients | | SAC |
| 55. | Safety | | Listing of epidermis thickness for psoriasis patients | | SAC |
| 56. | Safety | | Raw sas output of statistical analysis results for change from baseline LAG3+ and CD3+ for healthy volunteers (DTH subjects) | | SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 57. | Safety | | Raw sas output of statistical analysis results for change from baseline in cells in lesional biopsies measured by IHC for psoriasis patients | | SAC |
| 58. | Safety | | Raw sas output of statistical analysis results for change from baseline in epidermis thickness for psoriasis patients | | SAC |
| 59. | Safety | | Listing of sLAG-3 for healthy volunteers | | SAC |
| 60. | Safety | | Listing of sLAG-3 for psoriasis patients | | SAC |
| 61. | Safety | | Listing of blood transcriptomics for healthy volunteers | Includes raw Ct as well as average (mean delta Ct, delta delta Ct and fold change) | SAC |
| 62. | Safety | | Listing of blood transcriptomics for psoriasis patients | | SAC |
| 63. | Safety | | Listing of biopsy transcriptomics for psoriasis patients | | IA2 W2 |
| 8<br>1 | Safety | other | Listing of PPD challenge for healthy volunteers (DTH subjects) | | SAC |

# 14.10. Appendix 10: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request.